#### NCT05777174

#### CLINICAL STUDY PROTOCOL

An Open Label, Multi-Center, Safety and Pharmacokinetic Bridging Study of MB-102 (Relmapirazin) and the Use of the MediBeacon® Transdermal GFR Measurement System using the TGFR Reusable Sensor with Disposable Adhesive Ring in Normal and Renal Compromised Subjects for the Evaluation of Kidney Function

**Protocol Number:** 100-201

**Investigational Product:** MB-102 (Relmapirazin) / MediBeacon<sup>®</sup> Transdermal GFR

Measurement System

Phase: Bridging

**Sponsor:** MediBeacon Inc.

425 N. New Ballas Road St. Louis, MO 63141

**USA** 

**Date of Protocol** 2 April 2024

**Version of Protocol:** Version 5.1

#### **CONFIDENTIAL**

This protocol may not be reproduced or communicated to a third party without the written permission of MediBeacon Inc.

#### **Statement of Compliance**

The study will be conducted in compliance with the protocol, International Conference on Harmonization Good Clinical Practice E6 R2 (ICH-GCP), The Code of Federal Regulations Title 21 CFR Parts 812, 11, 50, 54 and 56 and ISO 14155: 2020 (3<sup>rd</sup> Edition) Clinical Investigation of Medical Devices for Human Subjects – Good Clinical Practice

# 1 Synopsis

| Protocol Number: | 100-201 |
|---|---|
| Title: | An Open Label, Multi-Center, Safety and Pharmacokinetic Bridging Study of MB-102 (Relmapirazin) and the Use of the MediBeacon® Transdermal GFR Measurement System using the TGFR Reusable Sensor with Disposable Adhesive Ring in Normal and Renal Compromised Subjects for the Evaluation of Kidney Function |
| Investigational | MB-102 (Relmapirazin) |
| Products: | MediBeacon® Transdermal GFR Measurement System (TGFR) |
| Number of Study<br>Sites: | This study will take place at up to 5 investigational sites in the US. |
| Phase: | Bridging |
| Objectives: | <ul> <li>To establish that the MB-102 transdermal fluorescence measured GFR using the MediBeacon<sup>®</sup> Transdermal GFR Measurement System with the TGFR reusable sensor with disposable adhesive ring is comparable to the measured MB-102 plasma GFR</li> <li>To evaluate the safety and effectiveness of the MediBeacon<sup>®</sup> Transdermal GFR Measurement System and the TGFR reusable sensor with disposable adhesive ring for the non-invasive transdermal fluorescence detection of MB-102 in subjects</li> </ul> |
| Study Design: | <ul> <li>Multi-center, bridging, adaptive open-label pharmacokinetic study comparing transdermal measured GFR (tGFR) to plasma-derived indexed GFR (nGFR).</li> <li>As the reusable sensor is new, an adaptive trial design will be employed.</li> <li>Run-in cohort of up to 30 evaluable subjects will commence the study. Additional Run-in subjects may be enrolled at new clinical sites to ensure protocol compliance. Run-in subject data will be considered tuning data.</li> <li>Validation Cohort 1 (approximately 20 evaluable subjects) will be used to confirm final algorithm selection. Validation Cohort 1 subject data will be considered tuning data.</li> <li>Validation Cohort 2 (approximately 75 evaluable subjects) will be analyzed in an interim analysis to compare results against the primary endpoint specification. If the primary endpoint has been achieved, the study will be terminated. If not, the trial will be continued.</li> <li>Validation Cohort 3 (approximately 65 evaluable subjects) will be enrolled in the event the interim analysis did not meet the primary outcome measure. Final analysis will be of the 140 evaluable subjects.</li> </ul> |
| Number of Treated<br>Subjects: | Up to 240 subjects are planned for enrollment. The population will be split into stratums in accordance with screening eGFR measured by the CKD-EPI equation (pre-2021): • Stratum 1: 50% of evaluable subjects with an eGFR ≥ 70 mL/min/1.73 m² • Stratum 2: 50% of evaluable subjects with an eGFR < 70 mL/min/1.73 m² Approximately 50% of subjects within each Stratum enrolled will be Fitzpatrick skin scale (FSS) I-III and 50% of subjects will have FSS IV-VI. Subjects will be |

| | enrolled across a spectrum of both eGFR (≤120 - ≥15 mL/min/1.73 m²) and FSS. An adaptive trial design will be employed. A Run-in cohort of 30 evaluable subjects and Validation Cohort 1 of up to 20 evaluable subjects with a mixture of eGFR and FSS will enroll to provide tuning data and allow algorithm finalization. This will be followed by up to 140 additional evaluable subjects enrolled: after 75 evaluable subjects in Validation 2 Cohort have been completed, an interim analysis will be conducted to compare results against the primary endpoint specification. If the primary endpoint has been achieved, the study will be terminated. If not, the trial will be continued with Validation Cohort 3 antil 140 evaluable subjects are enrolled. |
|---|---|
| | Subjects with incomplete assessments or major protocol deviations may be replaced. Thus, a maximum of 240 subjects may be enrolled. |
| Treatment: | Eligible subjects in stratums 1 and 2 will receive a single 130 mg dose of MB-102. Subjects who enroll in the Run-in and/or Validation 1 Cohort may repeat the study. Blood draws will be taken at pre-defined timepoints and the MediBeacon® Transdermal GFR Measurement System fluorescent measurements will be |
| C. I. D | collected over a 12 hour - 24 hour or longer period. |
| Study Duration per Subject: | Screening period: up to 28 days prior to dosing; dosing day, and a follow-up visit |
| Study Population: | within 7+/-3 days of dosing. Main Criteria for Inclusion: |
| | 1. Age ≥ 18 years – male or female a. Eligible female non-pregnant subjects who are either not of child-bearing potential or willing to use adequate contraception during the trial b. Males must be willing to practice abstinence or utilize adequate contraception from dosing day to at least 7 days post-dose c. For women of child-bearing potential, the subject should have a negative serum pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly i.e. abstinence, oral contraceptive either combined or progesterone alone; injectable progesterone, implants of levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, IUD device or system or male partner sterilization d. Men will not donate sperm during the study and for 1 month following the last dose of study drug 2. Subjects who are capable of directly providing informed consent and who can comply with the requirements and restrictions required by the protocol 3. Adequate venous access sufficient to allow blood sampling per protocol requirements Main Criteria for Exclusion: |
| | 1. Subjects positive for COVID-19 at the time of dosing |
| | 2. Recent donation or loss of blood or plasma: 100 mL to 499 mL |

| | within 30 days prior to the initial dose of the study medication; or more than 499 mL within 56 days prior to the initial dose of study medication 3. Non-steroidal anti-inflammatory (NSAID) use within 3 days of MB-102 dosing 4. The subject has participated in a clinical trial and has received an investigational product within the following time ranges: prior to the first dosing day in the current study: either 30 days or 5 half-lives of the investigational product (whichever duration is longer). 5. History of skin sensitivity to adhesives (e.g. Band-Aids, surgical tape) 6. History of severe allergic hypersensitivity reactions (unacceptable adverse events) or anaphylactoid reaction to any allergen including drugs, MB-102 or other related products (intolerance to a drug is not considered a drug allergy). 7. Any characteristics which, in the opinion of the investigator, makes the subject a poor candidate for participation in the clinical trial. 8. Significant scaring, tattoos or alterations in pigmentation on the sternum or other sensor location testing areas that would alter sensor readings versus other areas of the skin 9. Use of tanning sprays, tanning products etc. on the upper chest within 2 weeks of dosing day 10. Use make-up, lotions, Vaseline or other products on the area of the upper chest on the day prior to or the day of dosing 11. Any serious or uncontrolled medical disorder, active infection, physical exam finding, laboratory finding, or psychiatric condition that in the opinion of the investigator would limit the subjects' ability to complete study requirements or may put the subject at increased risk or compromise the interpretability of study results. 12. Currently receiving dialysis 13. Currently anuric 14. Subjects with positive serum pregnancy test 15. Subjects with an eGFR > 120 mL/min/1.73m <sup>2</sup> |
|---|---|
| Primary Endpoint: | The primary endpoint is the performance measure of P30 for transdermal-derived GFR with respect to the plasma-derived indexed GFR, with a 95% confidence interval. The performance goal is 85%. Success for the study will be that the lower limit of the 95% CI is greater than 85%. |
| Safety Evaluation | <ul> <li>Safety of MB-102 will be evaluated through treatment emergent adverse events (TEAEs), where treatment emergence is defined with respect to the first administration of MB-102.</li> <li>Safety of the MediBeacon® Transdermal GFR Measurement System will be evaluated through TEAEs, where treatment emergence is defined with respect to the start time of device use.</li> </ul> |

| Statistical Analyses | The primary endpoint is the performance measure of P30 for transdermal-derived GFR with respect to the plasma-derived indexed GFR, with a 95% confidence interval. The performance goal is 85%. Success for the study will be that the lower limit of the 95% CI is greater than 85%. Safety of MB-102 will be evaluated through treatment emergent adverse events (TEAEs), where treatment emergence is defined with respect to the administration of MB-102. Safety of the MediBeacon® Transdermal GFR Measurement System will be evaluated through TEAEs, where treatment emergence is defined with respect to the start time of Transdermal GFR Measurement System use. |
|---|---|
| | Additional safety variables include physical examinations, vital sign measurements, ECGs, clinical laboratory assessments, and medication use. |
| Sample Size | Prior data demonstrated for a P30 true value of 0.95, alpha of 0.025, |
| Determination | performance goal of 85%, power of 90%, the one-sided exact binomial test yields a sample size of 102. |
| Time Schedule: | Planned Start of Study: Q1 2023 |
| | Planned End of Study: Q2 2024 |

## **DOCUMENT APPROVALS**

Richard Dorshow, PhD President & Chief Scientific Officer

Joseph Pierro, MD Acting Head: Medical Affairs

Nancy Morrison Acting Head: Regulatory Affairs

Elizabeth LaPointe, MA Acting Head: Clinical Operations

# **Table of Contents**

| 1 | Syn | opsis | 2 |
|---|---|---|---|
| 2 | List | of Abbreviations and Definition of Terms | 10 |
| 3 | Int | oduction | 12 |
| 3 | 3.1 | Background | |
| | 3.2 | Nonclinical Data | |
| | 3.3 | Clinical Data | |
| | 3.4 | Study Rationale | |
| 4 | Stu | dy Objectives | 15 |
| 5 | Inv | estigational Plan | 15 |
| | 5.1 | Overall Study Design and Plan | |
| | <b>5.2</b> | Overview of Study Procedures | 16 |
| | 5.3 | Discussion of Study Design | 17 |
| | <b>5.4</b> | Selection of Study Population | 17 |
| | 5.4. | 1 Number of Planned Evaluable Subjects | 17 |
| | 5.4. | 2 Inclusion Criteria | 18 |
| | 5.4. | | |
| | 5.4. | r r r | |
| | 5.4. | 5 Replacement of Subjects | 19 |
| | 5.5 | Investigational Device | |
| | 5.5. | | |
| | 5.5. | | |
| | 5.5. | | |
| | 5.5. | 5 · | |
| | 5.5. | 5 Storage, Supply and Return/Destruction | 21 |
| | 5.5. | <b>y</b> | |
| | 5.6 | Investigational Drug | |
| | 5.6. | 7 0 | |
| | 5.6. | 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 3 | |
| | 5.6. | | |
| | 5.6. | | 24 |
| | 5.6. | | |
| | 5.7 | ${\bf Contact\ Procedures\ for\ Medical\ Issues\ Requiring\ Immediate\ Attention\}$ | |
| | 5.8 | Prior and Concomitant Therapy | |
| | 5.8. | | |
| | 5.8. | 2 Stable Use of Immunosuppressive Medications | 25 |
| 6 | Stu | dy Procedures | |
| | 6.1 | Schedule of Assessments and Procedures | |
| | 6.2 | Pre-screening | |
| | 6.3 | Screening | |
| | 6.4 | Night before Dosing Day | |
| | 6.5 | Dosing Day: Baseline Assessments | |
| | 6.6 | MB-102 Dosing | 31 |

| 6.7 | | |
|---|---|---|
| | 6.7.1 Stratum 1 (12 hour follow-up) | |
| 6.8 | | |
| 6.9 | · | |
| | 6.9.1 Sensor Cleaning | |
| | 6.9.2 Sensor Disinfection | |
| | 10 Follow-up Visit | |
| | 11 Early Withdrawal / Unscheduled Visits | |
| 6.3 | 12 Repeat Subjects | 36 |
| <b>7</b> ] | Efficacy and Safety Variables | 37 |
| | 1 Efficacy and Safety Measurements Assessed and Flow Chart | 37 |
| | 7.1.1 Efficacy Assessments | 37 |
| | 7.1.2 Safety Assessments | 37 |
| 7.2 | 2 Safety Review Committee | 44 |
| <b>8</b> | Information for the Investigator: Potential Risks of the Device | 4.4 |
| o 1<br>8.1 | | 44 |
| 8.2 | | |
| _ | 8.2.1 Adhesive Clip | |
| 8.3 | * | |
| | 8.3.1 Dose Extravasations | |
| | Statistical Methods | |
| 9.1 | | |
| 9.2 | · <b>/ F</b> | |
| 9.3 | , 1 | |
| 9.4 | · | |
| 9.5 | - J - F J | |
| 9.0 | | |
| | 9.6.1 Treatment-Emergent Adverse Events | |
| | 9.6.2 Physical Examinations/Limited Physical Assessments | |
| | 9.6.3 Clinical Laboratory Assessments | |
| | 9.6.4 ECGs | |
| | 9.6.5 Prior and Concomitant Therapies | |
| 9. | real | |
| 9.8 | 0 | |
| <b>10</b> | Quality Assurance and Quality Control | |
| 10 | • | |
| _ | 0.2 Audit and Inspection | |
| _ | 0.3 Monitoring | |
| | 0.4 Data Management and Coding | |
| | 0.5 Protocol Deviations | |
| 10 | 0.6 Direct Data Collection | 52 |
| 11 | Records / Retention | 52 |
| 12 | Ethics | 54 |

**15.2** 

| 12.1 | Independent Ethics Committee (IEC) | 54 |
|-------------------|------------------------------------------------|----|
| 12.2 | Ethical Conduct of the Study | |
| 12.3 | Subject Information and Consent | 54 |
| 12.4 | Financing and Insurance | |
| 12.5 | Subject Confidentiality | 55 |
| 12.6 | Reporting and Publication, Including Archiving | 55 |
| l3 Re | eferences | 56 |
| | ppendix A Fitzpatrick Scale | |
| l4 Aj | | 57 |
| l4 A <sub>l</sub> | ppendix A Fitzpatrick Scale | 57 |

Medical Officer ......59

## 2 List of Abbreviations and Definition of Terms

| AEI Acute kidney injury ALP Alkaline phosphatase ALT Alanine transaminase ALT Alanine transaminase AST Aspartate aminotransferase BMI Body Mass Index BP Blood pressure BUN Blood urea nitrogen CFR Code of Federal Regulations CKD Chronic kidney disease CKD-EPI Chronic kidney disease – epidemiology collaboration CO2 Carbon dioxide COVID-19 Coronavirus disease 2019 CRF Case report form CI Chloride Cr Creatinine CrCI Creatinine clearance CV Coefficient of variation ECG Electrocardiogram eCRF Electronic case report form EDC Electronic data capture EDC Electronic data capture EAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I lodine IB Investigator's Brochure ICF informed Consent Form ICH Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INN International Council on Harmonisation IV Intravenous K Potassium K, SEDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities MIIII National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Monus (OFFR) | | |
|---|---|---|
| ALP Alkaline phosphalase ALT Alanine transaminase AST Aspartate aminotransferase BMI Body Mass Index BP Blood pressure BUN Blood urea nitrogen CFR Code of Federal Regulations CKD Chronic kidney disease CKD-EPI Chronic kidney disease – epidemiology collaboration CO2 Carbon dioxide COVID-19 Coronavirus disease 2019 CRF Case report form Cl Chloride Cr Creatinine CrCl Creatinine CrCl Creatinine clearance CV Coefficient of variation ECG Electronic data capture eGFR Electronic data capture eGFR Electronic data capture eGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GIP Good Laboratory Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I lodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IP Investigational Device Exemption IV Intravenous K Potassium K2EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities ML Milliliter InGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | AE | |
| AST Aspartate aminortransferase BMI Body Mass Index BP Blood pressure BUN Blood urea nitrogen CFR Code of Federal Regulations CKD Chronic kidney disease – epidemiology collaboration CO <sub>2</sub> Carbon dioxide COVID-19 Coronavirus disease 2019 CRF Case report form CI Chloride Cr Creatinine CrCl Creatinine CrCl Creatinine CrCl Creatinine ECG Electrocardiogram eCRF Electronic case report form EDC Electronic data capture eGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GI.P Good Aboratory Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I lodine IB Investigator's Brochure ICF Indexpendent Ethics Committee INR International Council on Harmonisation ICU Intensive Care Unit INR INR International Organization for Standardization IV Intravenous K Potassium KzEDT A Potassium KzEDT A Potassium HAGDIANA Medical Dictionary for Regulatory Activities mIL Milliliter INGFR Indexpendent Ethics Committee INR INR International Organization for Standardization IV Intravenous IN Medical Dictionary for Regulatory Activities INR INH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | AKI | Acute kidney injury |
| AST BMI Body Mass Index BP Blood pressure BUN Blood urea nitrogen CFR Code of Federal Regulations CKD Chronic kidney disease CKD-EPI Chronic kidney disease – epidemiology collaboration CC <sub>0</sub> Carbon dioxide COVID-19 Coronavirus disease 2019 CRF Case report form CI Chloride Cr Creatinine CrCI Creatinine CCCC Creatinine clearance CV Coefficient of variation ECG Electroardiogram ECRF Electronic case report form EDC Electronic data capture EGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I lodine IB Investigator's Brochure ICC informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International Organization for Standardization IV Intravenous K Potassium K_SEDTA Potassium K_SEDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory drug OM Operational Manual | ALP | Alkaline phosphatase |
| BMI Blood pressure BUN Blood urea nitrogen CFR Code of Federal Regulations CKD Chronic kidney disease – epidemiology collaboration CO2 Carbon dioxide COVID-19 Coronavirus disease 2019 CRF Case report form CI Chloride Cr Creatinine CrCl Creatinine CrCl Creatinine CrCl Creatinine CFR Electronic case report form EDC Electrocardiogram eCRF Electronic case report form EDC Electronic data capture eGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I lodine IB Investigation's Brochure ICF informed Consent Form ICU Intensive Care Unit IDE Investigational Device Exemption IV International Organization for Standardization IV International Product ISO International Organization for Standardization IV Intravenous K Potassium K Pota | ALT | Alanine transaminase |
| BP Blood pressure BUN Blood urea nitrogen CFR Code of Federal Regulations CKD Chronic kidney disease CKD-EPI Chronic kidney disease – epidemiology collaboration CO2- Carbon dioxide COVID-19 Coronavirus disease 2019 CFF Case report form Cl Chloride Cr Creatinine CrCl Creatinine elearance CV Coefficient of variation ECG Electroardiogram eCRF Electronic case report form EDC Electronic data capture eGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Aboratory Practice GFR Glomerular filtration rate HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I I I I I I I I I I I I I I I I I I I | AST | Aspartate aminotransferase |
| BP Blood pressure BUN Blood urea nitrogen CFR Code of Federal Regulations CKD Chronic kidney disease CKD-EPI Chronic kidney disease – epidemiology collaboration CO2- Carbon dioxide COVID-19 Coronavirus disease 2019 CFF Case report form Cl Chloride Cr Creatinine CrCl Creatinine elearance CV Coefficient of variation ECG Electroardiogram eCRF Electronic case report form EDC Electronic data capture eGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Aboratory Practice GFR Glomerular filtration rate HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I I I I I I I I I I I I I I I I I I I | BMI | Body Mass Index |
| BUN Code of Federal Regulations CKD Chronic kidney disease CKD-EPI Chronic kidney disease – epidemiology collaboration CO2 Carbon dioxide COVID-19 Coronavirus disease 2019 CRF Case report form Cl Chloride Cr Creatinine CrCl Creatinine clearance CV Coefficient of variation ECG Electronic data capture eGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I I I I I IB Investigation's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IV Intravenous K Potassium K, Potassium K, Potassium K, Potassium MedDRA Medical Dictionary for Regulatory Activities mL Milliliter INGFR Indexed plasma glomerular filtration rate NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | BP | |
| CRD Chronic kidney disease CKD-EPI Chronic kidney disease — epidemiology collaboration CCD-EPI Chronic kidney disease — epidemiology collaboration COy Carbon dioxide COVID-19 Coronavirus disease 2019 CRF Case report form CI Chloride Cr Creatinine CrCl Creatinine clearance CV Coefficient of variation ECG Electrocardiogram eCRF Electronic case report form EDC Electronic data capture eGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I Iodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International Product INR International Product INR International Product ISO International Product INR International Product ISO International Product INR International Product ISO International Product INR International Product ISO International Product INR International Product INR International Product ISO International Product INR International Product ISO International Product ISO International Product INR INTERNATION Product INR INTERNATION Product INR INTERNATION Product INR INTERNATION Product | | • |
| CKD Chronic kidney disease CKD-EPI Chronic kidney disease – epidemiology collaboration CCo Co Carbon dioxide COVID-19 Coronavirus disease 2019 CRF Case report form Cl Chloride Cr Creatinine CrCl Creatinine clearance CV Coefficient of variation EGG Electrocardiogram eCRF Electronic data capture eGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GBP Good Manufacturing Practice GMP Good Manufacturing Practice GMP Good Manufacturing practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I I Iodine IB Investigation's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International Organization for Standardization IV Intravenous K Potassium K-EDDA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities ML Milliliter ING Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| CKD-EPI CO2 Carbon dioxide COVID-19 Coronavirus disease 2019 CRF Case report form Cl Chloride Cr Cr Creatinine CrCl Creatinine clearance CV Coefficient of variation ECG Electroardiogram eCRF Electronic case report form EDC Electronic data capture eGFR Electronic data capture EGFR Electronic data capture EGFR ESImated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP GGO GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I I lodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International Organization for Standardization IV Intravenous K K,2EDTA Potassium Hoskilliter InGFR Indexed plasma glomerular filtration rate NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| CO2 COVID-19 Coronavirus disease 2019 CRF Case report form Cl Chloride Cr Creatinine CrCl Creatinine CCCI Electronic data capture CGCR Electronic data capture CGFR Electronic data capture CGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration CGCP Good Clinical Practice GFR Glomerular filtration rate CGLP Good Laboratory Practice GMP Good Manufacturing Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT HEENT Head, Ears, Eyes, Neck, Throat I I I I I I I I I I I I I I I I I I I | | |
| COVID-19 Coronavirus disease 2019 CRF Case report form Cl Chloride Cr Creatinine CrCl Creatinine CrCl Creatinine CV Coefficient of variation ECG Electrocardiogram eCRF Electronic case report form EDC Electronic data capture eGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I lodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International Organization for Standardization IV Intravenous K Potassium K2EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory drug OM Operational Manual | | 1 01 |
| CRF Cl Chloride Cr Chloride Cr Creatinine CrCl Creatinine clearance CV Coefficient of variation ECG Electroacidogram eCRF Electronic case report form EDC Electronic data capture eGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I lodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International Product ISO International Organization for Standardization IV Intravenous K Potassium KzEDTA Potassium KzEDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory drug OM Operational Manual | | |
| CI Chloride Cr Creatinine CrCl Creatinine clearance CV Coefficient of variation ECG Electrocardiogram eCRF Electronic case report form EDC Electronic data capture eGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I Iodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International normalized ratio IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium KyEDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| Cr Creatinine CrCl Creatinine clearance CV Coefficient of variation ECG Electrocardiogram eCRF Electronic case report form EDC Electronic data capture eGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I I I I I I I I I I I I I I I I I I I | | • |
| CrCl Creatinine clearance CV Coefficient of variation ECG Electrocardiogram eCRF Electronic case report form EDC Electronic data capture eGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I lodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International Organization for Standardization IV Intravenous K Potassium K-EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory drug OM Operational Manual | | |
| CV Coefficient of variation ECG Electrocardiogram eCRF Electronic case report form EDC Electronic data capture eGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I lodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International Organization for Standardization IV Intravenous K Potassium KzEDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliture of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| ECG Electronic case report form EDC Electronic data capture eGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I Iodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International Product ISO International Organization for Standardization IV Intravenous K Potassium K2EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| eCRF Electronic case report form EDC Electronic data capture eGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I Iodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International Organization for Standardization IV Intravenous K Potassium KzEDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter INSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| EDC eGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I Iodine IB Investigator's Brochure ICF informed Consent Form ICH Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International Organization for Standardization IV Intravenous K Potassium K EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH NAtional Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| eGFR Estimated glomerular filtration rate FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I Iodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International normalized ratio IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium K_EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | • |
| FAS Full Analysis Set FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I Iodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International Organization for Standardization IV Intravenous K Potassium K2EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| FDA Food and Drug Administration GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I Iodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International normalized ratio IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium K <sub>2</sub> EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| GCP Good Clinical Practice GFR Glomerular filtration rate GLP Good Laboratory Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I Iodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International normalized ratio IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium K <sub>2</sub> EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | · |
| GFR GLP Good Laboratory Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I Iodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International normalized ratio IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium K <sub>2</sub> EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| GLP Good Laboratory Practice GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I Iodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International normalized ratio IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium K2EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| GMP Good Manufacturing Practice HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I Iodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International normalized ratio IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium K2EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| HCG Human chorionic gonadotropin HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I Iodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International normalized ratio IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium K2EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| HCT Hematocrit HEENT Head, Ears, Eyes, Neck, Throat I Iodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International normalized ratio IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium K2EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| HEENT Head, Ears, Eyes, Neck, Throat I Iodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International normalized ratio IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium K2EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities ML Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| I Iodine IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International normalized ratio IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium K2EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| IB Investigator's Brochure ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International normalized ratio IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium K2EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| ICF informed Consent Form ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International normalized ratio IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium K₂EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| ICH International Council on Harmonisation ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International normalized ratio IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium K2EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| ICU Intensive Care Unit IDE Investigational Device Exemption IEC Independent Ethics Committee INR International normalized ratio IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium K2EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| IDE Investigational Device Exemption IEC Independent Ethics Committee INR International normalized ratio IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium K2EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| IEC Independent Ethics Committee INR International normalized ratio IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium K2EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Millilter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| INR International normalized ratio IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium K <sub>2</sub> EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | • |
| IP Investigational Product ISO International Organization for Standardization IV Intravenous K Potassium K <sub>2</sub> EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| ISO International Organization for Standardization IV Intravenous K Potassium K <sub>2</sub> EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| IV Intravenous K Potassium K <sub>2</sub> EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | C C C C C C C C C C C C C C C C C C C |
| K Potassium K <sub>2</sub> EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | | |
| K <sub>2</sub> EDTA Potassium ethylenediaminetetraacetic acid MedDRA Medical Dictionary for Regulatory Activities mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | IV | |
| MedDRAMedical Dictionary for Regulatory ActivitiesmLMilliliternGFRIndexed plasma glomerular filtration rateNIHNational Institute of HealthNSAIDNon-steroidal anti-inflammatory drugOMOperational Manual | | |
| mL Milliliter nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | $K_2EDTA$ | Potassium ethylenediaminetetraacetic acid |
| nGFR Indexed plasma glomerular filtration rate NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | MedDRA | Medical Dictionary for Regulatory Activities |
| NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | mL | Milliliter |
| NIH National Institute of Health NSAID Non-steroidal anti-inflammatory drug OM Operational Manual | nGFR | Indexed plasma glomerular filtration rate |
| OM Operational Manual | NIH | |
| OM Operational Manual | NSAID | Non-steroidal anti-inflammatory drug |
| ORFM Optical Renal Function Monitor (now TGFR) | OM | Operational Manual |
| <u> </u> | ORFM | Optical Renal Function Monitor (now TGFR) |

| OTC | Over the counter |
|---------|------------------------------------------------|
| PA | Physical Assessment (limited) |
| PE | Physical exam (full) |
| PI | Principal Investigator |
| PK | Pharmacokinetic |
| POC | Point of care |
| PP | Per Protocol |
| RBC | Red blood cell |
| SAE | Serious Adverse Event |
| SAF | Safety Analysis Set |
| SAP | Statistical Analysis Plan |
| SCr | Serum creatinine |
| SNR | Signal to Noise Ratio |
| Tc-DTPA | Technetium diethylene triamine - pentaacetate |
| TEAE | Treatment-emergent adverse event |
| tGFR | Transdermal Glomerular Filtration Rate |
| TGFR | MediBeacon® Transdermal GFR Measurement System |
| UADE | Unanticipated Adverse Device Effect |
| Vd | Volume of Distribution |
| WBC | White blood cell |
| WHO | World Health Organization |
| WOCBP | Women of Child-Bearing Potential |

#### 3 Introduction

## 3.1 Background

Therapeutic interventions for acute kidney injury (AKI) patients are delayed due to current clinical practice of reliance on a serum creatinine blood test (SCr) for an estimation of glomerular filtration rate (GFR). Typically, 24-72 hours elapse from onset of a kidney injury event to a SCr indicating a non-normal level (Stevens et al, 2006). Since AKI affects upwards of 20% of hospitalized patients and 70% of critically ill patients in the intensive care unit (ICU), this contributes to high mortality rates (approaching 60% for those requiring renal replacement therapy [Endre at al., 2011]), development of chronic kidney disease (affecting an estimated 27 million Americans, accounting for ~ 24% of Medicare costs [NIH 2008]), and consequent progression to end stage renal disease (with an estimated 400,000 Americans on dialysis [Kidney Disease Statistics for the US]).

Glomerular filtration rate (GFR) is widely accepted as the best indicator of kidney function and is a key component of the diagnosis and management of renal impairment. A simple, accurate, and point-of-care (POC) method for determining GFR is needed, as current methods for determining GFR are either: 1) practical but lack accuracy, or 2) accurate but prohibitively complex, especially for frequent and recurrent measurements.

Current medical practice for general renal function assessment relies on estimated GFR (eGFR). This involves estimation using equations based on a single serum creatinine (SCr) measurement, or a measurement of creatinine clearance (CrCl) based on a 24-hour collection of urine plus measurement of a single SCr concentration. Although readily available and convenient, measurement of SCr as an indicator of renal function is problematic because it is a lagging indicator of current renal function, lacks sensitivity, and may be misleading because it is affected by age, state of hydration, renal perfusion, muscle mass, dietary intake, and many other anthropometric and clinical variables (Agarwal, 2003 and Verhave et al., 2005). CrCl estimation using timed urine collections can be more accurate, but problems with completeness of 24-hour urine collection often result in under or over estimation of CrCl.

Measuring GFR using urinary or plasma clearance of exogenous filtration markers is the accepted standard for evaluation of kidney function. In the past three decades, renally filtered exogenous agents such as inulin, iohexol, <sup>125</sup>Iodine-iothalamate (<sup>125</sup>I-iothalamate), and technetium-99m-diethylene triamine - pentaacetate (<sup>99m</sup>Tc-DTPA) have all been used to determine GFR (Stevens et al., 2006). From both a safety and effectiveness standpoint, these agents are acceptable, although they contain iodine, which can cause anaphylactoid reactions, and they can be nephrotoxic when very high volumes are used. However, they are not used routinely to determine GFR because the protocols are time-consuming, complex, and expensive, which make their repeated use impractical in many clinical settings, and they may require imaging equipment and administration of radioactive agents (Stevens and Levey, 2009). Accurate measurement of GFR at the patient's bedside is highly desirable in order to assess the patient's renal function. There is a significant need to develop a simple, accurate, and POC method for measuring GFR (Erley et al., 2001).

To address this unmet clinical need, MediBeacon is developing a combination product that requires the administration of a fluorescent tracer agent designated relmapirazin (also known as MB-102 and formerly known as MP-3180) that will be detected transdermally by a sensor which is attached to a device monitor (called the MediBeacon® Transdermal GFR Measurement System [TGFR]).

MB-102 has been engineered to be excreted from the body by the renal system, and specifically by the GFR mechanism. Normal functioning kidneys will remove this agent from the body with an approximate 2 hour half-life. Impaired functioning kidneys will take longer to excrete the agent and hence result in a longer half-life.

The sensor contains the light source for excitation of the tracer agent, the agent having a peak absorption wavelength of 440 nm. The detector is able to acquire the emission of the tracer agent, the agent having a peak emission wavelength of 560 nm. The sensor for the TGFR device is small and limited to the materials necessary for excitation and acquisition. Collection and processing of the data is performed within the monitor. The device monitor displays the TGFR data.

An initial algorithm had been developed from the Pilot 2 study data to convert measured fluorescence half-life data to GFR. Additional Pilot 2 study groups refined this algorithm for efficacy and robustness, as well as adding to the algorithm database. This algorithm was further tested in the Pivotal Trial 100-003 using the single use Brilliance sensor.

The TGFR reusable sensor with disposable adhesive ring is based off of the single use Brilliance sensor tested in protocol 100-003. This sensor is revised for serviceability by the end user for reuse of up to 100 times. The sensor base can be released by a clipping mechanism, facilitating easy reapplication of a new disposable adhesive ring. The sensor itself can be cleaned and disinfected between uses.

This sensor has the same light source, detector, and senses tracer and endogenous autofluorescence in the same way as the Brilliance sensor. The sensor interfaces and operates with the Brilliance monitor in the same manner as the original single use Brilliance sensor.

#### 3.2 Nonclinical Data

Available nonclinical study data on MB-102 support that the chemistry of the drug substance/drug product, and the manufacturing of the drug substance/drug product does not present a risk to human subjects. Additional information on the 29 nonclinical studies performed on MB-102 is found in the Investigator's Brochure.

#### 3.3 Clinical Data

A total of 586 subjects have been treated with an IV administration of MB-102 across the three pilot studies (Pilot 1A, Pilot 1B and Pilot 2 Groups 1, 2 and 3) and a completed Pivotal trial and including subjects enrolled in this trial as of the date of this protocol amendment. The Pilot 1

studies enrolled subjects with an eGFR indicating normal renal function. The Pilot 2 study and pivotal trial enrolled subjects with normal renal function and those with renal function in the CKD stage 1-5 range. In addition, a total of 22 subjects (11 healthy volunteers and 11 Crohn's patients) have received a 4 or 8 µmol/kg oral dose of MB-102 in a study evaluating the use of MB-102 in the evaluation of gut permeability (MediBeacon Protocol 300-01). The total population exposure to MB-102 as of this protocol is 608 subjects. A total of 95 subjects (16.0% of the total population across 6 studies) were reported to have adverse events (AE). All reported events were mild or moderate in severity. No severe events have been reported, nor have any serious adverse events been reported or unanticipated adverse device effects.

There have been no clinically significant findings with regard to vital signs, clinical laboratory results, physical exams or ECGs. Overall MB-102 administered intravenously at a dose of 4 μmol/kg whether or not followed by a 5 mL (milliliter) dose of iohexol (Omnipaque<sup>TM</sup> 300), or at a fixed dose of 130 mg / 7 mL (n=282) or consumed orally at a dose of 4 μmol/kg (n=8) or 8 μmol/kg (n=14) was well tolerated in the populations studied to date.

Adverse events related to the device itself were due to the adhesive materials used to hold the MediBeacon® Transdermal GFR Measurement System (TGFR) sensor in place. All device related events were considered mild or moderate in severity. For more information, please see the Investigator's Brochure.

MB-102 equilibrates between the vasculature and tissues post IV administration. The plasma pharmacokinetics show a peak concentration at the first sample time point. In Pilot 1A and Pilot 2, the first sample time point taken was approximately 5 minutes post administration; in Pilot 1B the first sample time point taken was approximately 30 minutes post administration. The fluorescence pharmacokinetics, reflecting the agent concentration in the tissue, has a peak fluorescence intensity in the range of 30 - 90 minutes, depending on the subject. MB-102 concentration equilibration between the vasculature and the tissue occurs approximately 30-60 minutes after the peak.

In the Pilot 2 Groups 1 and 2, the first blood draw was taken at 5 minutes post administration of MB-102, and the last at 12 hours post administration. The transdermal fluorescence was measured at the sternum and one other location for each subject using the prototype device QuantumLeap and Radiance. For all 140 subjects over the wide range of GFR values, the following were observed:

- A two-compartment plasma pharmacokinetic profile
- A high correlation between the MB-102 and iohexol plasma derived GFR values
- A high correlation between the MB-102 plasma and transdermal fluorescence pharmacokinetics

More information is available in the Investigator's Brochure.

#### 3.4 Study Rationale

This clinical study will evaluate the use of MB-102 and the MediBeacon® Transdermal GFR

2 April 2024 

Measurement System using the TGFR reusable sensor with disposable adhesive ring for the purpose of bridging the marketing application with a more useable sensor.

## 4 Study Objectives

The objectives of this pivotal study are:

- To establish that the MB-102 transdermal fluorescence measured GFR using the MediBeacon® Transdermal GFR Measurement System with the TGFR reusable sensor with disposable adhesive ring is comparable to the measured MB-102 plasma GFR
- To evaluate the safety and effectiveness of the MediBeacon® Transdermal GFR Measurement System with the TGFR reusable sensor with disposable adhesive ring for the non-invasive transdermal fluorescence detection of MB-102 in subjects

#### 5 Investigational Plan

## 5.1 Overall Study Design and Plan

Protocol 100-201 is a multi-center, open-label, adaptive bridging investigation studying the safety and pharmacokinetics of MB-102 and the use of the MediBeacon<sup>®</sup> Transdermal GFR Measurement System with the TGFR reusable sensor with disposable adhesive ring in normal and compromised renal function subjects with different skin color types comparing tGFR to plasma derived indexed GFR (nGFR).

Up to 240 subjects are planned to be dosed. The population will be split into stratums in accordance with eGFR by the CKD-EPI equation (pre- 2021) (Levey et al., 2009). The study will enroll into 4 consecutive cohorts:

1. A **Run-in Cohort** of up to 30 evaluable subjects will be enrolled to test monitor algorithm settings with the TGFR reusable sensor with disposable adhesive ring. Additional Run-in subjects may be enrolled at new clinical sites to ensure protocol compliance. Run-in subject data will be considered tuning data.

The following will be enrolled into the Run-in cohort:

- At least 5 subjects will be enrolled in Stratum 2
- At least 4 subjects in each of the FSS I-II: III-IV and V-VI

Clinical sites not yet active on the trial may also be required to participate in the Run-in Cohort in order to demonstrate protocol compliance prior to participating in the Validation 2 Cohort or Validation 3 Cohort.

- 2. **Validation Cohort 1** (approximately 20 evaluable subjects) will be used to confirm final algorithm selection. Validation Cohort 1 subject data will be considered tuning data.
- 3. **Validation Cohort 2** (approximately 75 evaluable subjects) will be analysed in an interim analysis to compare results against the primary endpoint specification. If the primary endpoint has been achieved, the study will be terminated. If not, the trial will be continued.

2 April 2024 

4. **Validation Cohort 3** (approximately 65 evaluable subjects) will be enrolled in the event the interim analysis did not meet the primary outcome measure. Final analysis will be of the 140 evaluable subjects.

Subjects will be screened, FSS determined by Mexameter, and if deemed eligible, will be enrolled. On treatment day, subjects will have the TGFR reusable sensor with disposable adhesive ring placed on their chest, and the MediBeacon® Transdermal GFR Measurement System will be initiated to collect background fluorescence. When this is completed, subjects will then receive a single dose of MB-102. Serial PK draws will be collected over a 12 or 24 hour (or longer) period (depending upon enrolment strata). Fluorescent measurements will also be collected during this period. For subjects with significant renal compromise, fluorescent measurements will continue until the sensor no longer detects MB-102 in the body. Following completion of the monitoring period, subjects will return to the study center approximately 1 week later for a safety follow-up visit.

Subjects who do not complete the study or considered not evaluable (major protocol deviations, extravasations, etc.) may be replaced. Up to 240 total subjects may be enrolled.

## **5.2** Overview of Study Procedures

Potential subjects will be screened for eligibility within 28 days prior to planned dosing. Based on their screening eGFR (measured using the CKD-EPI equation), they will be assigned to Stratum 1 or Stratum 2:

- Stratum 1: eGFR  $\geq$  70 mL/min/1.73 m<sup>2</sup> (50% of subjects)
- Stratum 2: eGFR <  $70 \text{ mL/min/1.73 m}^2 (50\% \text{ of subjects})$

Following pre-dose procedures to ensure eligibility, one sensor will be affixed to the subject on the upper chest in the area between the shoulders (including the pectoralis and sternum area). The subject will then receive the MB-102 injection. MB-102 will be administered by IV injection over 30-60 seconds, followed by a saline flush IV over 30-60 seconds.

Stratum 1: PK sampling will be collected pre-dose and at 5, 15, 30, 60, 90, 120, 180, 240, 300, 360, 480, 600 and 720 minutes post-dose (12 hour collection period).

Stratum 2: PK sampling will be collected pre-dose and at 5, 15, 30, 60, 90, 120, 180, 240, 300, 360, 480, 600, 720 960, 1200, and 1440, minutes post-dose (24 hour collection period).

Safety assessments in the form of vital signs, safety labs, ECGs, and adverse event collection will occur during the dosing day.

Within 7 +/- 3 days of dosing, subjects will return to the study center for additional safety follow-up assessments.

2 April 2024 

## 5.3 Discussion of Study Design

The study is designed to validate the performance of the TGFR Measurement System using the TGFR reusable sensor with disposable adhesive ring.

## 5.4 Selection of Study Population

## 5.4.1 Number of Planned Evaluable Subjects

The study may enroll up to 240 subjects across 4 consecutive cohorts in order to obtain 140 evaluable subjects. Unevaluable subjects are those with major protocol deviations that impact efficacy (such as no reported average session tGFR, premature sensor removal, extravasations, etc.). The cohorts include:

- 1. Run-in Cohort (approximately 30 subjects)
- 2. Validation Cohort 1 (approximately 20 subjects)
- 3. Validation Cohort 2 (approximately 75 evaluable subjects)
- 4. Validation Cohort 3 (approximately 65 evaluable subjects)

After 75 evaluable subjects in the Validation 2 Cohort have been completed, an interim analysis will be conducted to compare results against the primary endpoint specification. If the primary endpoint has been achieved, the study will be terminated. If not, the trial will continue with enrolment into Validation Cohort 3 until 140 evaluable subjects are enrolled.

The population will be split into stratums in accordance with eGFR by the CKD-EPI equation (pre-2021):

- Stratum 1: 50% of subjects with an eGFR  $\geq$  70 mL/min/1.73 m<sup>2</sup>
- Stratum 2: 50% of subjects with an eGFR  $< 70 \text{ mL/min/1.73 m}^2$

Subjects will be targeted across the spectrum of eGFR from normal through Stage 4 CKD. Subjects with an eGFR > 120 mL/min/1.73 m<sup>2</sup> or < 15 mL/min/1.73 m<sup>2</sup> will be excluded. Efforts will be made to balance enrollment across the following eGFR levels such that each subcategory has at least 6 subjects enrolled:

- $\geq 90 \leq 120 \text{ mL/min}/1.73 \text{ m}^2$
- $\overline{60} 89 \text{ mL/min/1.73 m}^2$
- $45 59 \text{ mL/min}/1.73 \text{ m}^2$
- $30 44 \text{ mL/min/1.73 m}^2$
- $15 29 \text{ mL/min/1.73 m}^2$

Approximately 50% of subjects within each stratum enrolled in the US will be Fitzpatrick Skin Scale (FSS) I-III and 50% of subjects will have FSS IV-VI. Subjects will be targeted across the full spectrum of FSS (I-VI) such that FSS cohorts I-II, III-IV and V-VI will each enroll no less than 6 subjects.

#### **5.4.2** Inclusion Criteria

To be eligible for study entry, all subjects must satisfy all of the following criteria:

#### **Main Criteria for Inclusion:**

- 1. Age  $\geq$  18 years male or female
  - a. Eligible female non-pregnant subjects who are either not of child-bearing potential or willing to use adequate contraception during the trial
  - b. Males must be willing to practice abstinence or utilize adequate contraception from dosing day to at least 7 days post-dose
  - c. For women of child-bearing potential, the subject should have a negative serum pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly i.e. abstinence, oral contraceptive either combined or progesterone alone; injectable progesterone, implants of levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, IUD device or system or male partner sterilization
  - d. Men will not donate sperm during the study and for 1 month following the last dose of study drug
- 2. Subjects who are capable of directly providing informed consent and who can comply with the requirements and restrictions required by the protocol
- 3. Adequate venous access sufficient to allow blood sampling per protocol requirements

#### **5.4.3** Exclusion Criteria

To be eligible for the study, subjects must not meet any of the criteria noted below:

- 1. Subjects positive for COVID-19 at the time of dosing
- 2. Recent donation or loss of blood or plasma: 100 mL to 499 mL within 30 days prior to the initial dose of the study medication; or more than 499 mL within 56 days prior to the initial dose of study medication
- 3. Non-steroidal anti-inflammatory (NSAID) use within 3 days of MB-102 dosing
- 4. The subject has participated in a clinical trial and has received an investigational product within the following time ranges: prior to the first dosing day in the current study: either 30 days or 5 half-lives of the investigational product (whichever duration is longer).
- 5. History of skin sensitivity to adhesives (e.g. Band-Aids, surgical tape)
- 6. History of severe allergic hypersensitivity reactions (unacceptable adverse events) or anaphylactoid reaction to any allergen including drugs, MB-102 or other related products (*intolerance to a drug is not considered a drug allergy*).
- 7. Any characteristics which, in the opinion of the investigator, makes the subject a poor candidate for participation in the clinical trial
- 8. Significant scaring, tattoos or alterations in pigmentation on the sternum or other sensor location testing areas that would alter sensor readings versus other areas of the skin

2 April 2024 

- 9. Use of tanning sprays, tanning products etc. on the upper chest within 2 weeks of dosing day
- 10. Use make-up, lotions, Vaseline or other products on the area of the upper chest on the day prior to or the day of dosing
- 11. Any serious or uncontrolled medical disorder, active infection, physical exam finding, laboratory finding, or psychiatric condition that in the opinion of the investigator would limit the subjects' ability to complete study requirements or may put the subject at increased risk or compromise the interpretability of study results.
- 12. Currently receiving dialysis
- 13. Currently anuric
- 14. Positive serum pregnancy test
- 15. Subjects with an eGFR > 120 mL/min/1.73m<sup>2</sup>

#### 5.4.4 Removal of Subjects from Therapy or Assessments

In accordance with applicable regulations, a subject has the right to withdraw from the study at any time and for any reason without prejudice to his or her future medical care by the investigator or at the institution where the subject's care is provided.

Reasons for withdrawal from the study may include one or more of the following:

- Withdrawal of consent
- Administrative decision by the PI or MediBeacon
- Adverse event requiring removal from the study
- Physician prescribes a treatment that would conflict with the subject's continued participation in the study

Subjects withdrawing from the study will be encouraged to complete the follow-up study visit including all safety evaluations. The reason(s) for withdrawal will be documented.

Reasonable efforts will be made to contact subjects who are lost to follow-up. All attempts and contacts must be documented in the subject's file.

The sponsor has the right to terminate the study at any time due to a safety issue or if special circumstances arise making further treatment of subjects impossible. In this event, the investigator(s) will be informed of the reason for study termination.

## 5.4.5 Replacement of Subjects

Should a subject meet eligibility, but is unable to be scheduled for dosing, that subject will be considered a screen failure. In addition, subjects who are unable to have a tGFR measured by the MediBeacon® TGFR Measurement System (due to premature sensor removal, for example) or a major protocol deviation (such as a dosing extravasation) may be replaced to ensure the minimum evaluable sample size is enrolled. All subjects with exposure to MB-102 will be included in the safety analysis.

2 April 2024 

### 5.5 Investigational Device

MediBeacon<sup>®</sup> Transdermal GFR Measurement System (TGFR) is an investigational device that is intended to measure the Glomerular Filtration Rate (GFR) in patients with normal or impaired renal function by noninvasively monitoring fluorescent light emission from an exogenous tracer agent (MB-102) over time.

Site staff will place and affix the TGFR reusable sensor and disposable adhesive ring for all enrolled subjects. One sensor will be attached to the upper chest. An adhesive clip, surgical tape or other means may also be used to alleviate tension on the sensor cord. Additional instructions for sensor placement will be provided in the Study Procedure Manual.

The TGFR reusable sensor and disposable adhesive ring is revised for serviceability by the end user for reuse of up to 100 times. The sensor base can be released by a clipping mechanism, facilitating easy reapplication of a new disposable adhesive ring.

The sensor itself must be cleaned and sanitized between uses. To clean, the sensor is wiped with a damp cloth wetted with a mild detergent mixed with a 20:1 ratio of water to detergent. To sanitize, the sensor should be wiped with a 70% alcohol wipe or an equivalent lint free wipe wetted with a 70% isopropyl alcohol solution. This sensor has the same light source, detector, and senses tracer and endogenous autofluorescence in the same way as the Brilliance sensor. The sensor interfaces and operates with the Brilliance monitor in the same manner as the Brilliance sensor.

The only parts of the MediBeacon® TGFR reusable sensor and disposable adhesive ring that come into contact with the subject are the single-use adhesive pad, and the optical window. The optical window protrudes very slightly from the adhesive, ensuring consistent contact with the subject's skin. The self-adhesive pad is similar to those used for disposable ECG patches. The sensor remains affixed to the subject for at least 12.5 hours for Stratum 1 and up to or exceeding 24 hours for Stratum 2 subjects.

#### 5.5.1 Premature Dislodgment of a TGFR Sensor from the Skin

Should a sensor be prematurely dislodged from the subject's skin during the measurement period and after injection with MB-102, it will not be replaced and the subject will be discontinued from the measurement period of the study (but will remain in the trial to be followed for safety). End of treatment assessments should be collected (safety labs, vitals, and ECG). If a sensor dislodges from the skin during the baseline period (prior to MB-102 injection), a new sensor may be used and the study re-started.

The TGFR is designed to require a clean baseline (pre-injection of MB-102) in order to accurately measure GFR. If MB-102 is in the body at the time a sensor is attached, it will not allow measurement.

#### **5.5.2** Sensor Detachment from the TGFR Monitor

If a sensor becomes detached even temporarily from the TGFR monitor, there will be loss of data for the period of time until the sensor is reattached. The sensor should be re-plugged into the monitor and the prompts on the screen should be followed so that fluorescent measurements can continue. This occurrence should be recorded as a major protocol deviation if the tGFR is NOT reported, and a minor deviation if the monitor displays the tGFR.

## **5.5.3** Identity of Investigational Device

The MediBeacon<sup>®</sup> Transdermal GFR Measurement System is manufactured by MediBeacon Inc. (St. Louis, MO, USA). All packaging and labeling operations will be performed according to current Good Manufacturing Practice (GMP), ISO 13485 and the relevant regulatory requirements.

## 5.5.4 Labeling

Each MediBeacon<sup>®</sup> Transdermal GFR Measurement System monitor and each sensor will be clearly labelled with a Serial Number and REF MDB (Rev).

Each device will be labelled with the following information:

## CAUTION

Investigational Device.
Limited by United States
Law to Investigational Use.

Additional labels will include the following information:

REF MDB ###### Rev 0# LOT MDBNNNNNN-## SN. ####### Non Sterile

## 5.5.5 Storage, Supply and Return/Destruction

Multiple investigational devices (monitors and sensors) will be provided to the clinical sites. Disposable items (disposable sensor ring and adhesive materials) will be single-subject use only. Devices and disposable materials must be stored in a secure location and are only for use during the clinical trial. All devices will be returned to the Sponsor at the conclusion of the trial. Instructions for return will be included in the Study Procedure Manual.

### **5.5.6** Device Accountability

All inventory received for clinical trial use will be tracked. All inventory will be returned to MediBeacon or disposed of following instructions from the Sponsor. An investigational device accountability record will be kept current and will contain:

- Subject ID (screening number)
- Device(s) monitor serial number
- Sensor serial number
- Date of dosing
- Any observations noted during the use of the device

## 5.6 Investigational Drug

MB-102 (relmapirazin) is a bis-serine aminopyrazine that will be used as an exogenous fluorescent Glomerular Filtration Rate (GFR) agent. This agent is excited by blue light and emits green light.

MB-102 has the following characteristics:

- Produces fluorescence in vivo when excited by blue light, which can be reliably detected by transdermal measurement when MB-102 is injected intravenously
- Has elimination kinetics that allows determination of GFR from fluorescence measurement within a clinically useful timeframe
- Is filtered by the kidney
- Is not protein bound
- Is not expected to undergo secretion or tubular reabsorption
- Is not expected to be metabolized by the liver or other organs
- Is not expected to affect kidney function
- Has been shown to be safe in animal models, in therapeutic dose range
- Is photostable in its administration form and during sample handling and analysis
- Has been shown to be a GFR tracer agent in nonclinical animal models and early clinical studies

#### 5.6.1 Stability of Drug Product

### **5.6.1.1** Active Pharmaceutical Ingredient (API)

A sixty (60) month stability-testing program conducted under Good Manufacturing Practices (GMP) for the Active Pharmaceutical Ingredient (API) Lot # 07-130227-02/02-43-01 (140 grams manufactured April 2013 by Cambrex Inc., formerly PharmaCore) used in the Pilot 1 and 2 studies was completed. Stability conditions was  $25^{\circ}\text{C} \pm 2^{\circ}\text{C}$ ,  $60\% \pm 5\%$  R.H. Results at 60 months show negligible degradation in active ingredient purity and essentially no change in the total impurity amount with respect to the zero time parameters.

A sixty (60) month stability-testing program conducted under GMP for a second API lot (1 kg manufactured in August 2017 by Cambrex), API Lot # 2337-1706-00256 is on-going. Stability conditions was  $25^{\circ}\text{C} \pm 2^{\circ}\text{C}$ ,  $60\% \pm 5\%$  R.H. Results show negligible degradation in active ingredient purity and essentially no change in the total impurity amount with respect to the zero time parameters at the five year (and final) time point.

A third GMP API lot of 1 kg was manufactured in June 2020 by Cambrex, Lot # 2337-2004-00667. A sixty (60) month stability-testing program has been initiated and is ongoing at conditions of  $25^{\circ}\text{C} \pm 2^{\circ}\text{C}$ ,  $60\% \pm 5\%$  R.H. Results show negligible degradation in active ingredient purity and essentially no change in the total impurity amount with respect to the zero time parameters at the three year time point.

Three batches of API have been manufactured at the commercial manufacturing facility (Regis Technologies) and stability has been initiated and is on-going. Results for all three lots (including Lot M20213-980-11) show negligible degradation in active ingredient purity and essentially no change in the total purity amount with respect to the zero-time parameters at the twelve-month time point.

The samples for long term stability testing of registration Lots M24213-980-11, M24218-975-9, and M24241-978-6 were stored at 25°C  $\pm$  2°C, 60% R.H.  $\pm$  5%, relative humidity and accelerated stability stored at 40°C  $\pm$  2°C, 75% R.H.  $\pm$  5%.

#### **5.6.1.2** Formulated Product

A 12 month stability-testing program for the GMP formulated product Batch P02213 (~1500 mL), manufactured in April 2013 by AMRI (formerly Aptuit) from API Lot # 07-130227-02/02-43-01, which was used for the Pilot 1A and 1B studies, has been completed. Results show negligible degradation in active ingredient purity and essentially no change in the total impurity amount with respect to the zero time parameters for the 2 - 8°C condition.

A 24 month stability-testing program for the GMP formulated product Batch P03915 (~3200 mL), manufactured in May 2015 by AMRI from API Lot # 07-130227-02/02-43-01, and which was used for Groups 1 and 2 in Protocol ORFM Pilot 2 study, has been completed. Stability condition was 2 - 8°C. Results show negligible degradation in active ingredient purity and essentially no change in the total impurity amount with respect to the zero time parameters.

Formulated product with designation Batch P04517 (~9000 mL) was manufactured under GMP conditions by AMRI using API Lot # 2337-1706-00256. This batch was placed on stability at 2 - 8°C for a three year period. At the 36 month time point, there was negligible degradation in active ingredient purity and essentially no change in the total impurity amount.

Stability testing of the GMP formulated product Batch MLF001 (registration batch manufactured by Curia in Albuquerque, New Mexico) from drug substance batch M24213-980-11 evaluated physical, chemical, and microbiological attributes at designated time points. At the nine month

2 April 2024 

time point, all samples (upright and inverted) stored at the  $5^{\circ}\text{C} \pm 3^{\circ}\text{C}$  storage conditions have met specifications.

#### 5.6.2 Identity of Investigational Drug

MB-102 is packaged in amber vials at a concentration of 18.6 mg/mL in a 7.4 mL volume. MB-102 in formulation includes the following: sodium dihydrogen phosphate monohydrate, sodium hydroxide, sodium chloride, water for injection. Instructions for preparation of MB-102 will be included in the Study Procedure Manual.

#### 5.6.3 Investigational Drug Labeling

MB-102 drug labels for US distribution include the following information:

Relmapirazin

7 mL of MB-102 Solution for injection only 18.6 mg/mL

Lot No: MLF001

Mfg. Date: 06/15/2022 Store at 2°C - 8°C

Caution: New Drug – Limited by Federal (United States) law to Investigational use.

Manufactured for MediBeacon

#### 5.6.4 Investigational Drug Storage, Supply, Return/Destruction

Relmapirazin vials should be stored at  $2^{\circ}C - 8^{\circ}C$  in a secure location. Temperature records will be maintained by the clinical site.

All study medications will be stored, reconciled and either returned to the sponsor or destroyed according to applicable regulations following authorization by MediBeacon.

#### 5.6.5 Investigational Drug Accountability

Drug accountability will be maintained by the clinical site and will be reviewed during the study and 100% reconciled at the conclusion of the trial.

Drug accountability documentation may include, but may not be limited to, the following information:

- Receipt date
- Lot
- Expiry and/or manufacture date
- Dispensing information

## 5.7 Contact Procedures for Medical Issues Requiring Immediate Attention

Any medical-related issues or questions requiring immediate resolution or direction should be directed to the Sponsor medical monitor using the contact information listed below:

| Joseph | Pierro, | MD ( | Unit | ted | States) |
|--------|---------|------|------|-----|---------|
| Cell: | | | | | |
| Email: | | | | | |

For submission of Serious Adverse Event information or Unanticipated Adverse Device Effects, the following email maybe used:

• Email: Safety@medibeacon.com

#### 5.8 Prior and Concomitant Therapy

Throughout the study, investigators may prescribe concomitant medications or treatments deemed necessary to provide adequate care, with the exception of other investigational agents or drugs that may alter renal function. All attempts should be made to maintain the subjects on a stable dosing regimen of medications from screening through the duration of the study.

Concomitant medication information will be collected for all subjects within 3 days of dosing through the follow-up visit. Additionally, use of any non-drug procedural therapies will be recorded for each subject including the nature of the therapy, the date/time of the procedure, and the reason for the therapy. Concomitant medication information taken at the time of an SAE will also be collected during the safety data follow-up.

#### **5.8.1** Prohibited Concomitant Medications

The use of NSAIDs are prohibited 3 days prior to dosing for all subjects with the exception of low-dose (81 mg or less) aspirin.

## 5.8.2 Stable Use of Immunosuppressive Medications

The protocol currently allows for subjects on immunosuppressant medications. Those medications that fall into this category are found in **Table 1.** This table also outlines timelines around stability of those medications required at the time of dosing.

Table 1 Dose Stability Timelines for Subjects on Immunosuppressive Agents

| Immunosuppressive Agent | Dose Stability Timeframe |
|---------------------------------|---------------------------|
| Antithymocyte Globulin (rabbit) | No changes within 90 days |
| Basiliximab | No changes within 90 days |
| Infliximab | No changes within 90 days |
| Antithymocyte Globulin (equine) | No changes within 90 days |
| Rituximab | No changes within 90 days |
| Cyclosporine | No changes within 30 days |
| Tacrolimus | No changes within 30 days |

## **6 Study Procedures**

## 6.1 Schedule of Assessments and Procedures

The schedule of planned study assessments is shown in **Table 2.** 

**Table 2 Study Schedule of Events** 

| Period | Pre-Screen (optional) | Screening | Dosing Day | Dosing Day | Dosing Day | Dosing Day | Follow-up Visit |
|---|---|---|---|---|---|---|---|
| | | 28 days to day -2<br>prior to Dosing | Pre-dose | Dosing<br>(time 0) | During 12 – 24<br>hours post IP<br>injection | Completion of 12 hours<br>or up to 24 hours post<br>IP injection | 7 days +/- 3 days |
| Informed Consent <sup>a</sup> | X | X | | | | | |
| Inclusion / Exclusion | | X | X | | | | |
| Demographics | | X | | | | | |
| Medical History | | X | X | | | | |
| Pregnancy Test for WOCBP <sup>b</sup> | | X | X | | | | |
| PE or Limited PA <sup>c</sup> | | X | X | | | | X |
| Vital Signs <sup>d</sup> | | X | X | | X | X | X |
| Height and Weight <sup>e</sup> | | X | X | | | | |
| Clinical Labs <sup>f</sup> | | X | X | | | X | X |
| Mexameter measurements | X | X | X | | | | |
| Transdermal Data Collection <sup>g</sup> | | | X | X | X | X | |
| Drink water h | | | X | X | | | |
| Administration of MB-102 <sup>i</sup> | | | | X | | | |
| PK blood collection <sup>j</sup> | | | X | | X | X | |
| ECG <sup>k</sup> | | X | X | | | X | |
| Concomitant Therapies <sup>1</sup> | | X | X | | X | X | X |
| Adverse Events <sup>m</sup> | | | X | X | X | X | X |
| Document Fitzpatrick Skin<br>Color Type <sup>n</sup> | X | X | | | | | |

#### **Table 2 Legend**

- a. Pre-screening consent may be used to evaluate skin color only using the Mexameter device. Full informed consent is required prior to any study related procedures being conducted.
- b. Negative pregnancy serum human chorionic gonadotropin (hCG) test at screening for women of childbearing potential (WOCBP) is required for eligibility. On dosing day, a urine pregnancy test will be conducted for WOCBP who agree to use an acceptable method of birth control
- c. A full physical examination (PE) is required at the screening visit. A full PE or limited physical assessment (PA) will be conducted prior to dosing. (Limited PA includes assessments of HEENT, respiratory, cardiovascular, abdominal systems). A full or limited exam will be conducted at the follow-up visit.
- d. Vital signs include blood pressure, respiration rate, pulse and temperature. Note: temperature is collected at screening, pre-dose, at approximately 12 hours post-dose and at the follow-up visit (and not during multiple timepoints on dosing day). Whenever possible, the subject should be resting for approximately 5 minutes prior to all measurements. Vital signs will be collected at screening, pre-dose and at the following post-dose timepoints: 90, 250 and 500, 710 minutes (±5 min). For subjects followed for 24 hours, an additional measurement will be taken at 1450 minutes.
- e. Height and Weight should be measured at screening; height and weight will also be measured on the day of dosing.
- f. Clinical laboratory assessments will be analyzed by a central laboratory and consist of standard chemistry, hematology and urinalysis parameters per **Table 3.** Coagulation panel will be conducted at Screening only.
- g. MediBeacon<sup>®</sup> Transdermal GFR Measurement System baseline data collection will commence prior to dose administration. At least 15 minutes prior to dosing, sensors should be placed on the subject and the MediBeacon<sup>®</sup> Transdermal GFR Measurement System started. Data collection will continue through 12 24 hours of PK sampling. Once an tGFR is measured, sensors may be removed while PK sampling continues.
- h. The subject should be given 240 mL of ambient water to drink the night prior (if brought in the night before dosing), the morning of dosing, and just prior to MB-102 dose administration
- i. MB-102 will be administered as a dose of 130 mg (7 mL) via IV injection over a 30 60 second injection period. This will be followed by a saline flush over 30 60 seconds. Time of administration will be recorded.
- j. Stratum 1: PK sampling will be collected pre-dose and at 5, 15, 30, 60, 90 (±2 min), 120, 180, 240, 300, 360, 480, 600 and 720 (±5 min) minutes post-dose (12 hour collection period). Stratum 2: PK sampling will be collected pre-dose and at 5, 15, 30, 60, 90 (±2 min), 120, 180, 240, 300, 360, 480, 600, 720, 960, 1200, and 1440 (±5 min) minutes post-dose (24 hour collection period). Blood draws should be via a venous catheter and will be processed in accordance with instructions available in the Study Procedure Manual.
- k. A 12 lead ECG will be performed at Screening, prior to dosing, and at 700 minutes post dosing (±5 min). Subjects should be resting quietly for 10-15 minutes prior to the ECG collection.
- 1. Concomitant medications administered within 3 days prior to baseline through the final follow-up visit will be recorded.
- m. Adverse events are collected from the time of sensor placement (for baseline measurement) through the follow-up visit.
- n. Fitzpatrick Skin Scale will be assessed by evaluating the skin on the upper chest (where sensors will be placed) using the Mexameter measurement.

## 6.2 Pre-screening

US sites will have the option to pre-screen study subjects to evaluate them directly for skin color in order to meet Fitzpatrick Skin Scale stratification recruitment requirements. The Mexameter will be used to determine FSS type.

## 6.3 Screening

Screening will occur within 28 days (but at least 2 days prior to) the baseline / dosing day and will comprise of the following:

- Obtain written informed consent before any study-specific assessments are performed
- Assess eligibility against the inclusion and exclusion criteria
- Collect demographic data and medical history; review concomitant medications
- Obtain screening non-fasting laboratory tests including chemistry, hematology, and coagulation profile (See Section 7.1.2.6 and Table 3). Perform serum pregnancy test in women of child-bearing potential and collect a urine sample for urinalysis.
- Perform COVID-19 testing
- Collect height and weight measurements; ensure subjects are not wearing shoes
- Perform a full physical exam and collect vital signs including temperature (Sections 7.1.2.7 and 7.1.2.8)
- Perform a 12 lead ECG (Section 7.1.2.9)
- Document Fitzpatrick Skin Scale (FSS) Color Type by examining the upper chest (locations for possible sensor placement)) and perform Mexameter measurements to determine the FSS. Collect 3 melanin and erythema measurements to obtain an average value and use the following to determine the FSS value:

| 0 | FSS type I: | Mexameter melanin range: | 0 - 100 |
|---|---------------|--------------------------|-----------|
| 0 | FSS type II: | Mexameter melanin range: | 100 - 150 |
| 0 | FSS type III: | Mexameter melanin range: | 150 - 250 |
| 0 | FSS type IV: | Mexameter melanin range: | 250 - 350 |
| 0 | FSS type V: | Mexameter melanin range: | 350-450 |
| 0 | FSS type VI: | Mexameter melanin range: | 450 - 999 |

## 6.4 Night before Dosing Day

For institutions that prefer to bring study subjects to the institution the night before dosing day, the following procedures may be performed:

- Perform COVID testing
- Review subject eligibility
- Update medical history with any new information or issues since screening
- Perform a limited physical assessment
- Record concomitant medications taken within 3 days prior to dosing day
- Perform a urine pregnancy test for WOCBP
- Have the subject consume 240 mL of ambient water

## 6.5 Dosing Day: Baseline Assessments

Baseline assessments will be performed prior to dosing (with the exception of those procedures noted in Section 6.3 that were performed the night before for those sites that bring subjects in the night prior to dosing).

- Update medical history with any new information or issues occurring since the initial screening visit (if not performed the night before).
- Collect the subject weight and height (BSA and BMI will be calculated based on dosing day height and baseline weight measurements). Ensure subjects are not wearing shoes and only light clothing.
- Review subject eligibility
- Confirm that the subject has consumed 240 mL of ambient temperature water at least 1 hour prior to dosing time.
- Perform a limited physical assessment and collect vital signs (including temperature) (Sections 7.1.2.7 and 7.1.2.8).
- Perform a baseline ECG (Section 7.1.2.9).
- Record concomitant medications taken within 3 days of the dosing visit
- For WOCBP, a urine pregnancy test will be performed
- Clean and prepare the body areas for sensor attachment using an alcohol pad. Excess hair should be clipped (not shaved) from the area for sensor.
- Calibrate the Mexameter prior to use in accordance with instructions in the Study Procedure Manual. Record calibration results.

- Obtain melanin and erythema measurements with the Mexameter at the location of sensor placement (Section 7.1.2.11). Measurements should be reviewed, and the values should be within range of each other. Measurements with significantly disparate values should
- A venous catheter should be placed in one arm for PK blood draws. A pre-dose baseline draw should be collected.

be repeated as it is likely the probe position was on different locations on the body.

- Obtain baseline laboratory tests including chemistry, hematology, and urinalysis (See Section 7.1.2.6 and Table 3).
- Prior to dosing, confirm the sensor has been cleaned and disinfected (see Section 6.9). The device sensor should be attached to the subject and the MediBeacon® Transdermal GFR Measurement System data acquisition initiated. During this data acquisition period, no other study procedures should be performed and the subject should be asked to remain very still. This period requires approximately 20 30 minutes.
- Adverse event collection begins
- Prior to dosing, have the subject consume an additional 240 mL of ambient water
- Place a venous catheter for the purpose of MB-102 dosing in the opposite arm. An appropriately sized angio-catheter should be selected based on study subject (22 24 gauge is strongly recommended).
  - NOTE: The Sponsor may request that the placement of the dosing catheter occur BEFORE the sensor is attached to the subject. In these cases, the dosing catheter will be in place during the baseline data acquisition. The subject should be instructed to keep the arm with the dosing catheter very still, and the site should dose as quickly as possible after the "Administer Lumitrace" screen appears on the TGFR monitor.
  - o If the catheter is placed AFTER the baseline assessment is completed, sites should minimize the time between catheter placement and dosing to no more than 5 minutes. As catheter placement can be difficult in older subjects, if this duration exceeds 5 minutes, it should not be considered a protocol deviation.

#### **6.6** MB-102 Dosing

The dose of 130 mg MB-102 (7.0 mL injection) should be prepared based on instructions provided in the Study Procedure Manual. Final dose calculation should be based on weight and not volume, therefore dosing syringes will be weighed prior to administration. The prepared syringe should be maintained at ambient temperature. MB-102 dosing will be performed in the opposite arm from PK draws whenever feasible.

Administration of MB-102 will be via direct intravenous (IV) injection following angio-catheter placement. Care should be taken to prevent extravasations during dosing. Ideally, a 22-24-

V 5.1

gauge angio-catheter and 10 mL syringe should be used for administration. Catheter size will be collected.

- Ensure Universal Standard precautions are taken with handwashing and gloving procedures; maintain aseptic technique when handling the prepared syringe
- Check the patency of the placed catheter by injecting a small volume of saline prior to MB-102 dosing
- Administration of MB-102 should be via a steady IV injection (without hard pressure) over 30 60 seconds (smaller bore catheters [24 gauge] may require a slower injection)
- Following MB-102, a 10 mL saline flush should be administered over 30 60 seconds
- The injection site should be observed for swelling or induration or yellow discoloration indicative of a drug infiltration. Drug infiltration may also cause discomfort or pain to the study subject.
- The dosing catheter will be removed after the saline flush is completed.

To avoid extravasation/infiltration:

- Ensure no dislodgement of the needle cannula during venepuncture
- Ensure the back vein wall is not punctured during placement
- Avoid strong pressure on the syringe plunger during saline or MB-102 administration
- Perform a slow injection over the full 30 60 seconds.

If an extravasation occurs, record it as both an adverse event and a protocol deviation. Subjects with evidence of MB-102 or saline extravasations will be discontinued from PK collection and fluorescent measurements but followed for safety. Subjects may be replaced at the discretion of the Sponsor.

The time noted at the start of MB-102 injection (but prior to the saline flush) is the start-time for the timing of the PK draws.

Following dosing, the syringe will be weighed in order to calculate an accurate dose of MB-102.

### **6.7** Post-dose Study Procedures

## 6.7.1 Stratum 1 (12 hour follow-up)

During the course of the study day, it is particularly important for site teams to check the patency of PK catheters. If a catheter is determined to be compromised in anyway, another catheter may be placed in the same arm as the original catheter utilizing a different vein. Direct sticks may also be used to obtain blood

PK draws will be drawn via the venous catheter at the following timepoints:

- PK draw in  $K_2$  EDTA tube at 5 minutes ( $\pm 2$  minute)
- PK draw in  $K_2$  EDTA tube at 15 minutes ( $\pm 2$  minute)

- PK draw in K<sub>2</sub> EDTA tube at 30 minutes (±2 minutes)
- PK draw in K<sub>2</sub> EDTA tube at 60 minutes (±2 minutes)
- PK draw in K<sub>2</sub> EDTA tube at 90 minutes (±2 minute)
- Vital sign collection at 90 minutes (±5 minutes)
- PK draw in  $K_2$  EDTA tube at 120 minutes ( $\pm 5$  minutes)
- PK draw in K<sub>2</sub> EDTA tube at 180 minutes (±5 minutes)
- PK draw in K<sub>2</sub> EDTA tube at 240 minutes (±5 minutes)
- Vital sign collection at 250 minutes (±5 minutes)
- PK draw in K<sub>2</sub> EDTA tube at 300 minutes (±5 minutes)
- PK draw in K<sub>2</sub> EDTA tube at 360 minutes (±5 minutes)
- PK draw in K<sub>2</sub> EDTA tube at 480 minutes (±5 minutes)
- Vital sign collection at 500 minutes (±5 minutes)
- PK draw in K<sub>2</sub> EDTA tube at 600 minutes (±5 minutes)
- Perform a 12 lead ECG at 700 minutes (±5 minutes)
- Vital sign collection (includes temperature) at 710 minutes ( $\pm 5$  minutes)
- PK draw in K<sub>2</sub> EDTA tube at 720 minutes (±5 minutes)
- Obtain laboratory tests including chemistry, hematology, and urinalysis (See Section 7.1.2.6 and Table 3) at 725 minutes (-245 minutes)
- At the conclusion of TGFR measurements (when tGFR is reported on the monitor), the sensor may be removed
- Adverse events will be collected based on subject reports and medical team observations

## 6.8 Stratum 2 (24 hour follow-up)

PK draws will be drawn via the venous catheter at the following timepoints:

- PK draw in  $K_2$  EDTA tube at 5 minutes ( $\pm 2$  minute)
- PK draw in K<sub>2</sub> EDTA tube at 15 minutes (±2 minutes)

- PK draw in K<sub>2</sub> EDTA tube at 30 minutes (±2 minutes)
- PK draw in  $K_2$  EDTA tube at 60 minutes ( $\pm 2$  minutes)
- PK draw in  $K_2$  EDTA tube at 90 minutes ( $\pm 2$  minute)
- Vital sign collection at 90 minutes (±5 minutes)
- PK draw in K<sub>2</sub> EDTA tube at 120 minutes (±5 minutes)
- PK draw in K<sub>2</sub> EDTA tube at 180 minutes (±5 minutes)
- PK draw in K<sub>2</sub> EDTA tube at 240 minutes (±5 minutes)
- Vital sign collection at 250 minutes (±5 minutes)
- PK draw in K<sub>2</sub> EDTA tube at 300 minutes (±5 minutes)
- PK draw in K<sub>2</sub> EDTA tube at 360 minutes (±5 minutes)
- PK draw in K<sub>2</sub> EDTA tube at 480 minutes (±5 minutes)
- Vital sign collection at 500 minutes (±5 minutes)
- PK draw in K<sub>2</sub> EDTA tube at 600 minutes (±5 minutes)
- Perform a 12 lead ECG at 700 minutes (±5 minutes)
- Vital sign collection (includes temperature) at 710 minutes (±5 minutes)
- PK draw in K<sub>2</sub> EDTA tube at 720 minutes (±5 minutes)
- Obtain laboratory tests including chemistry, hematology, and urinalysis (See Section 7.1.2.6 and Table 3) at 725 minutes (-245 minutes)
- PK draw in K<sub>2</sub> EDTA tube at 960 minutes (±5 minutes)
- PK draw in K<sub>2</sub> EDTA tube at 1200 minutes (±5 minute)
- PK draw in K<sub>2</sub> EDTA tube at 1440 minutes (±5 minutes)
- Vital sign collection at 1450 minutes (±5 minutes)
- At the conclusion of TGFR measurements (when an tGFR is reported on the monitor), the sensor may be removed.
- Adverse events will be collected based on subject reports and medical team observations

• Subjects may be discharged from the study center

## 6.9 Sensor Cleaning and Disinfection

Following removal of the sensor of the subject, the sensor must be cleaned and disinfected prior to use on subsequent subjects. A cleaning kit will be provided to the sites which will include a mild dish soap (detergent) and lint free cloths.

## 6.9.1 Sensor Cleaning

Sites will make a solution of 20:1 ratio of water to detergent. This mixture should not exceed 55°C (130°F).

Clean the surfaces of the TGFR Reusable Sensor with a damp cloth using 20:1 detergent mixture, removing all visible soil. Ensure all excess fluid is squeezed from the cloth before cleaning. If the cloth is excessively wet, the detergent and water solution may penetrate the sensor and affect functionality. After cleaning the TGFR Reusable Sensor, wipe the TGFR Reusable Sensor with a clean lint free damp cloth to remove the mild detergent mixture. Dry the TGFR Reusable Sensor with a clean lint free cloth. Never use an abrasive pad or abrasive cleaner on the monitor.

#### 6.9.2 Sensor Disinfection

The TGFR Reusable Sensor will be disinfected by wiping the surface with a 70% isopropyl alcohol wipe, or an equivalent lint free wipe wetted with 70% isopropyl alcohol. Wipe the TGFR Reusable Sensor as necessary to maintain visual wetness for a minimum duration of 2 minutes. After disinfecting the TGFR Reusable Sensor, allow each to air dry completely.

Sensor cleaning and disinfection will be documented on a log and maintained with the Investigator Site Files.

Caution: The use of other cleaners and disinfectants may cause significant damage to the TGFR Reusable Sensor and may impair its future use. Never use an abrasive pad on any surface of the TGFR sensor. Do not use Bleach or other solutions aside from what is described above. The TGFR Reusable Sensor is not designed to be immersed, soaked, rinsed, or sprayed with water. Do not immerse, soak, rinse, or spray the TGFR Reusable Sensor in water or other cleaning solutions. Failure to follow the cleaning procedures described herein could result in hazards to users, patients, and clinicians. As with any medical electrical equipment, care must be taken to prevent liquid from entering the TGFR Reusable Sensor to avoid electrical shock hazard, fire hazard, or damage to the electrical components.

#### 6.10 Follow-up Visit

Subjects will return for a safety follow-up visit approximately 7 +/-3 days after the dosing visit. The following assessments will be performed

- Perform a full or limited physical exam and collect vital signs including temperature (Sections 7.1.2.7 and 7.1.2.8)
- Obtain laboratory tests including chemistry, hematology, and urinalysis (Section 7.1.2.6 and Table 3).
- Record concomitant medications
- Collect adverse events; review ongoing AEs and document resolution (when applicable)

#### 6.11 Early Withdrawal / Unscheduled Visits

Any subject that withdraws from the study early for any reason, or who needs to have an unscheduled visit performed to assess a safety issue, will have the following assessments performed:

- Obtain laboratory tests including chemistry, hematology, and urinalysis profile (Section 7.1.2.6 and Table 3).
- Perform a full or limited physical exam and collect vital signs (Sections 7.1.2.7 and 7.1.2.8)
- Record concomitant medications
- Collect adverse events; review ongoing AEs and document resolution (when applicable)
- Record withdrawal date and reason for withdrawal, if appropriate

#### 6.12 Repeat Subjects

Subjects may be re-enrolled in the protocol in the following situations (and if no documented safety concerns regarding exposure to the investigational device or drug):

- If they were part of the Run-in Cohort and/or Validation Cohort 1
- When a dose extravasation has occurred
- When there is a device malfunction (sensor falling off during the monitoring period and before a tGFR has been reported)
- If no tGFR is reported due to another issue
- Back-up subjects who were not dosed

Stratum 1 subjects must have a minimum of a 3-day wash-out from prior exposure of MB-102 before receiving another dose. Stratum 2 subjects must have a minimum of a 5-day wash-out from prior exposure of MB-102 before receiving another dose.
In some cases, the screening visit (if outside the 28-day window) may need to be repeated. Repeat subjects enrolled into Validation Cohort 2 or 3 will be provided with a new subject ID, however the original subject ID will be cross-referenced in the database.

Subjects can be in the study a maximum of four times and only when the above situations have occurred. Subjects who successfully complete Validation Cohort 2 with full PK and an average session TGFR cannot repeat the study.

## 7 Efficacy and Safety Variables

## 7.1 Efficacy and Safety Measurements Assessed and Flow Chart

**Table 2** shows the planned study assessments.

#### 7.1.1 Efficacy Assessments

This bridging study is not designed to address treatment efficacy rather it is to evaluate the use of MB-102 and the MediBeacon® Transdermal GFR Measurement System using the TGFR resusable sensor and disposable adhesive ring to provide a point of care (POC) means to collect GFR data. The specific endpoints related to calculation of GFR are discussed in Section 9.

#### 7.1.2 Safety Assessments

Safety will be monitored by the assessments described below as well as the collection of AEs at every visit after screening. Planned safety assessments are detailed in the MediBeacon® Transdermal GFR Measurement System Study Schedule (**Table 2**). The investigators or site staff will be responsible for monitoring the safety of subjects who have entered this study and will be responsible for detecting, documenting and reporting events that meet the definition of an adverse event (AE) or serious adverse event (SAE). Significant findings that were noted to be present at or prior to dosing must be included in the relevant medical history page of the eCRF. Significant new findings that begin or worsen after dosing must be recorded on the AE page of the eCRF. Subjects should be followed until the event is resolved or stabilized. AEs are collected from the time of initial sensor placement until the completion of the follow-up visit.

#### 7.1.2.1 Adverse Events

#### **Adverse Event Definition**

An adverse event is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, temporally associated with the use of a medicinal product, whether or not related to the investigational medical device or drug.

An unanticipated adverse device effect (UADE) is any serious adverse effect on health or safety, any life-threatening problem or death caused by, or associated with a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the application; or any other unanticipated serious problem associated with a device that relates to

the rights, safety, or welfare of subjects. For the purposes of this trial, the device is the MediBeacon<sup>®</sup> Transdermal GFR Measurement System and the sensor system including the disposable adhesive ring for the attachment of the optical sensors to the body.

## **Documentation and Reporting of Adverse Events**

AEs should be reported and documented in accordance with the procedures outlined below. The following data should be documented for each AE:

- Description/term of the symptom event (underlying diagnosis)
- Date of first occurrence and date of resolution (if applicable)
- Classification of "serious" or "not serious" (Section 7.1.2.2)
- Severity
- Causal relationship
- Action taken
- Outcome of event

For abnormal clinically significant laboratory findings, the clinical manifestation (diagnosis) should be noted as an adverse event (e.g. anemia instead of low hemoglobin). Should a clinically significant lab abnormality occur that is not part of a diagnosis, the abnormality itself may be reported as an AE. Laboratory abnormalities that meet the criteria for an AE should be followed until they have returned to normal or an adequate explanation of the abnormality is determined. When an abnormal laboratory result corresponds to a sign/symptom of an already reported AE it is not necessary to separately record the lab result as an additional AE.

## **Assessment of Severity**

Each AE will be assigned a category by the investigator as follows:

- <u>Mild:</u> results in minimal transient impairment of a body function or damage to a body structure and/or does not require any intervention other than monitoring or OTC medication.
- Moderate: Results in moderate transient impairment of a body function or transient damage to a body structure and/or requires intervention, such as administration of medication or transfusion or laparoscopic or endoscopic procedure to prevent permanent impairment of a body function or damage to a body structure.
- <u>Severe:</u> An event which is life threatening, results in permanent impairment of a body function or permanent damage to a body structure or necessitates significant intervention, such as major surgery, to prevent permanent impairment of a body function or permanent damage to a body structure. The term severe is often used to describe the intensity (severity) of a specific event (as in mild, moderate, or severe myocardial infarction); the event itself, however, may be of relatively minor medical significance (such as severe

headache). This is not the same as serious, which is based on patient/event outcome or action criteria usually associated with events that pose a threat to a patient's life or functioning. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations. An event that changes in severity (gets worse or gets better) should be noted as its worst severity.

## **Assessment of Causality**

Every effort will be made by the investigator to assess the relationship of the AE, if any, to the study device (and components), investigational drug. Causality should be assessed using the categories presented below:

| TT 1 . 1 | O1: 1 | | 1 1 | 1 . 1 | , 1 1 . |
|---|---|---|---|---|---|
| Unrelated | ( linical event | t with an inco | mnatihle time | relationship to | o study device or |
| Omerated | Cilincal Cycii | t with an inco | mbanbie mine | TCIauonsino v | o study device of |

study drug, and that could be explained by underlying disease or other

drugs or is incontrovertibly not related to the study device.

Unlikely Clinical event whose time relationship to study device investigational

drug makes a causal connection improbable, but that could plausibly be

explained by underlying disease or other drugs.

Possible Clinical event with a reasonable time relationship to study device or

investigational drug, but that could also be explained by concurrent

disease or other drugs.

Probable Clinical event with a reasonable time relationship to study device or

investigational drug and is unlikely to be attributed to concurrent disease

or other drugs.

Very Likely/Certain Clinical event with plausible time relationship to study device or

investigational drug, and that cannot be explained by concurrent disease

or other drugs.

AEs that are deemed related should be further assessed to determine if a relationship to the investigational drug, or device can be elucidated.

#### **Action Taken**

The investigator will describe the action taken in the appropriate section of the eCRF, as follows:

- None
- Concomitant interventional treatment(s) administered (includes medications or procedures)
- Other, specify

#### **Outcome of the Event**

The investigator will describe the outcome of the event in the appropriate section of the eCRF, as follows:

Unknown

V 5 1

- Resolved
- Ongoing
- Resolved with sequelae
- Death (with date and cause reported)

## Follow-up of Adverse Events

Subjects with AEs should be followed until the event is resolved or until, in the opinion of the investigator and medical monitor, the event is stabilized or determined to be chronic.

#### 7.1.2.2 Serious Adverse Events

#### **Serious Adverse Event Definition**

An SAE is any AE from this study that results in one of the following outcomes:

An adverse event that:

- a) led to death;
- b) led to serious deterioration in the health or the subject, that either resulted in:
  - 1) a life threatening illness or injury or
  - 2) a permanent impairment of a body structure or a body function, or
  - 3) in-patient or prolonged hospitalization, or
  - 4) medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function;
- c) led to fetal distress, fetal death or a congenital abnormality or birth defect

Reporting requirements for all SAEs is detailed in Section 7.1.2.3.

Note: Planned hospitalization for a pre-existing condition, or a procedure required by the protocol without serious deterioration in health, is not considered a serious adverse event.

## 7.1.2.3 Reporting of Serious Adverse Events

Any SAE must be reported by the investigator if it occurs during the clinical study whether or not the event is considered to be related to the MediBeacon® Transdermal GFR Measurement System, or the investigational drug. All serious adverse events must be reported by the Investigator (or designee) by submitting the Serious Adverse Event Report Form (via the electronic data capture (EDC) system) or via email to MediBeacon within 24 hours of learning of the adverse event.

The Sponsor safety team, in cooperation with the Investigator, will assess all serious adverse events considered drug or device-related for potential reportability to regulatory authorities and ethical committees as an Unanticipated Adverse Device Effect (UADE) or as an expedited serious adverse event.

V 5 1

Note: It is also the responsibility of the Investigator to inform their Independent Ethics Committee (IEC) of other serious adverse events (i.e. non-UADEs) as required by their IEC procedures and in conformance with regulations.

# SAEs must be reported within 24 hours of knowledge.

For submission of Serious Adverse Event information or Unanticipated Adverse Device Effects, the following email maybe used:

Email: Safety@medibeacon.com

The investigator should not wait to receive additional information to document fully the event before notification to the Sponsor of an SAE, though additional information may be requested. Where applicable, information from relevant laboratory results, hospital case records, and autopsy reports should be obtained.

Instances of death, congenital abnormality, or an event that is of such clinical concern as to influence the overall assessment of safety, if brought to the attention of the investigator at any time and linked by the investigator to this study, should be reported to MediBeacon.

The sponsor or designee will promptly notify all relevant investigators and the regulatory authorities of findings that could adversely affect the safety of subjects, impact on the conduct of the study or alter the IEC approval/favorable opinion of the study. In addition, the sponsor, will expedite the reporting to all concerned investigators, to the IECs, and to the regulatory authorities of all adverse device reactions that are both serious and unanticipated.

#### 7.1.2.4 Pregnancies

Testing for pregnancy for a female study subject with childbearing potential must be conducted at screening (or within 7 days of dosing). In addition, a urine pregnancy test will be performed prior to dosing on treatment day. Subjects who are pregnant or intend to become pregnant during the study will be excluded. Should a pregnancy occur with a study subject, the pregnancy should be reported to MediBeacon within 24 hours of the site's knowledge. All pregnancies will be followed to term, delivery or premature termination.

#### 7.1.2.5 Device Observations / Malfunctions

All device observations, malfunctions or failures of the MediBeacon<sup>®</sup> Transdermal GFR Measurement System will be documented in the eCRF. In addition, failures of the sensor adhesive will be specifically documented.

## 7.1.2.5.1 Sensor Displacement

Prior dosing with MB-102:

Should a sensor be accidently removed (or significantly bumped) prior to administration of MB-102, it should be removed from the subject, the disposable ring removed and a new ring put on

the sensor and re-attached after re-cleaning the area with an ethanol wipe. Baseline measurements may then be re-started.

## After dosing with MB-102:

If a sensor is accidently removed (or significantly bumped) following administration of MB-102 but before a tGFR is calculated, the subject will remain in the study for safety follow-ups only for the full duration required by their stratum (12 hours or 24 hours). PK sample collection and fluorescent measurements will be terminated; however, safety assessments (vital signs, ECGs and clinical safety labs) will continue to be performed.

## 7.1.2.6 Clinical Laboratory Evaluation

Clinical laboratory assessments (**Table 3**) will be performed by a central lab. Reference ranges will be used by the investigator to assess the laboratory data for clinical significance and changes relative to baseline measurements. Clinically significant changes in laboratory values will be documented as adverse events.

**Table 3 Clinical Laboratory Analytes** 

| Chemistry Panel | Hematology | Other required lab tests |
|---|---|---|
| <ul> <li>Alkaline Phosphatase</li> <li>Alanine Aminotransferase (ALT)</li> <li>Albumin</li> <li>Aspartate Aminotransferase (AST)</li> <li>Bilirubin (total and direct)</li> <li>Blood Urea Nitrogen (BUN)</li> <li>Calcium (Ca)</li> <li>Carbon dioxide (CO2)</li> <li>Chloride (C)</li> <li>Creatinine (SCr)</li> <li>Glucose</li> <li>Phosphorus</li> <li>Potassium</li> <li>Sodium</li> <li>Total Protein</li> <li>Uric acid</li> <li>BUN/Creatinine ratio</li> </ul> All lab tests are non-fasting | <ul> <li>Hematology</li> <li>Hematocrit</li> <li>Hemoglobin</li> <li>WBC</li> <li>RBC</li> <li>Platelets</li> <li>Differentials</li> <li>Neutrophils</li> <li>Lymphocytes</li> <li>Monocytes</li> <li>Eosinophils</li> <li>Basophils</li> </ul> Coagulation Parameters <ul> <li>Only performed</li> <li>at screening</li> <li>PT</li> <li>INR</li> <li>aPTT</li> </ul> | For WOCBP Serum pregnancy test (screening and a urine dipstick on day of dosing Urinalysis Protein Glucose Ketones Hemoglobin Bilirubin Urobilinogen Acetone Nitrite Leucocytes pH Specific gravity Color Bacteria If abnormalities are seen, then microscopic examination will be performed |
| COVID-19 Test at screening and prior to dosing (local testing) | | |

# 7.1.2.7 Vital Signs

Vital signs (including blood pressure, pulse, respiration, and temperature) will be measured at screening, at multiple timepoints on dosing day(s), and at the follow-up visit. Vital signs should be collected while the subject is in a seated position and after resting for approximately 5 minutes for all measurements. Temperature is only collected at screening, pre-dose, and the completion of the dosing day, and at the follow-up visit.

## 7.1.2.8 Physical Examinations or Limited Physical Assessments

Physical examinations (when conducted by a physician, or other medically qualified investigator) or limited physical assessments (when performed by a nurse or other qualified individual) should include at a minimum an assessment of the head, ears, eyes, nose, throat (HEENT), respiratory, cardiovascular, and gastrointestinal systems. It is preferred that the same medical professional perform the baseline and post dosing assessments. Significant findings that were present prior to dosing must be included in the Medical History eCRF page. Significant new findings that begin or worsen after dosing must be recorded on the AE page of the eCRF. Clinically significant abnormalities occurring post-dose should be evaluated by a physician and noted as AEs.

The study investigator will assess the subject for the occurrence of clinically significant new findings that begin or worsen after dosing which must be recorded as an AE on the eCRF page. A full physical exam should be conducted at screening and limited physical assessments may be conducted at other time points and must also be inclusive of the relevant organ or body system of interest for assessing the AE.

#### 7.1.2.9 ECGs

Standard 12 lead ECGs will be collected at screening, prior to dosing and at 700 minutes (±5 min). The following parameters will be assessed: interpretation, ventricular rate, PR interval, QRS duration, QT, and QTcF.

Subjects should be allowed to rest quietly approximately 10-15 minutes prior to their ECG. Additional ECGs may be collected if an issue or safety concern is noted.

An appropriately trained and experienced investigator will interpret the ECGs. A subject with an abnormal clinically significant ECG during screening does not qualify for the study. A subject with an abnormal not clinically significant ECG does not qualify for dosing without investigator comment on the ECG source document/eCRF.

#### 7.1.2.10 PK Sample Collection

PK samples will be collected at the timepoints noted in **Table 2.** Recommendations for venous access and sample processing information are available in the Study Procedure Manual. PK samples should be collected in a manner to prevent haemolysis and placed on ice until processed and aliquoted into cryovials. PK samples must be stored frozen at -70 to -80°C until shipped for PK analysis.

#### 7.1.2.11 Mexameter® Measurements

A commercially available Mexameter<sup>®</sup> device will be provided to the sites for the measurement of skin pigment (melanin) and erythema. The device should be used in accordance with the instructions provided in the Study Procedure Manual (including pre-use calibration). Measurements should be performed on subjects when they are not in close proximity to a window and should be made on the approximate location of sensor placement. It is advisable, when required, to clip excess hair as early in the dosing day as possible to allow transient redness due to the clipping process to fade. The site should note any skin irritation due to clipping as medical history. Mexameter<sup>®</sup> measurements of melanin and erythema will be collected prior to sensor placement.

#### 7.2 Safety Review Committee

A Safety Review Committee (SRC) will be convened and will include the medical monitor, the safety manager(s), clinical monitor(s) and clinical manager. The SRC will oversee safety data (AEs, vitals, clinical labs, ECG data, etc.) generated by enrolled study subjects on the trial. In addition, they will review all SAEs and UADEs and clinically significant safety observations noted during the study. Oversight work and study related decisions will be performed in accordance with a written Safety Review Committee Plan.

#### 8 Information for the Investigator: Potential Risks of the Device

Adverse events that may be anticipated in this clinical study are outlined for the investigational drug and the MediBeacon® Transdermal GFR Measurement System.

#### 8.1 Investigational Drug

Clinical data from the Pilot 1A and 1B studies (total n = 32 subjects) included the following adverse events:

- Pilot 1A (n = 16)
  - Vasovagal reaction (1 subject)
  - o Dizziness (1 subject, 2 events)

These events occurred in fasting subjects shortly after dosing and resolved on that day. No other AEs, injection site reactions, clinically significant laboratory values or significant changes in vital signs were noted during this study.

- Pilot 1B (n = 16)
  - o Headaches (56.3% of subjects)
  - o Erythema (at the site of the adhesive) (100% of subjects)
  - o Diarrhoea (1 subject)
  - o Dizziness (occurring in 1 subject following release from the study center)

Erythema was thought to be related to the adhesive used to adhere the sensor to the skin. Headaches were deemed related to the head strap required to hold the forehead sensor in place. Sensor placement on forehead was discontinued post Pilot 1B.

MB-102 is excreted in the urine. Therefore, urine discoloration (chromaturia) is expected but has not been considered an adverse event in prior studies.

In the Pilot 2 study, a total of 234 subjects with normal to compromised renal function have been exposed to MB-102. A total of 120 subjects received a dose of 4 µmol/kg followed by a 5 mL injection of iohexol. Seventy (70) subjects received a single dose only (no iohexol) of 4 µmol/kg of MB-102) and 44 have received a fixed dose of 130 mg (7 mL). All reported AEs were mild or moderate in severity and resolved without sequalae. Overall, MB-102 given in conjunction with or without iohexol was well tolerated in this subject population.

A total of 40 adverse events were reported in 28 treated subjects in Groups 1, 2 and 3 for an AE rate of 12.0% in the treated population. A total of 31 events were considered mild and 9 moderate events occurred in 5 subjects (2.5% of the population). There were no severe events reported. There were no Serious Adverse Events (SAEs) reported during the study. There were no Unanticipated Adverse Device Effects (UADEs) reported during the study.

Four AEs, dyspepsia, chromaturia, hot flush and (facial) rash were considered related to investigational product (MB-102); all events resolved by study completion. Dyspepsia and chromaturia were also considered to be related to iohexol. Of note, chromaturia is an expected effect of MB-102 (noted in the Investigator's Brochure) and expected in all subjects as the excretion of MB-102 will color the urine of subjects receiving the product. It is not a documented effect of iohexol (per the label).

Seven (7) AEs occurring in 7 subjects were considered related to the device (sensor attachment); these included application site erythema, dermatitis, and pruritus and were considered related to the adhesive material used to hold the sensor in place. Two events of application site discoloration (melanin spot at the sensor location) were noted in 2 subjects in the SOG cohort which resolved within 24 hours of removal of the sensor. Other reported AEs (conjunctivitis, nausea, vomiting, cardiac murmur, headache, anxiety, micturition urgency, pollakiuria, urine odor abnormal, peripheral oedema, fatigue, and a pruritis event [not at the sensor location] were considered not related to MB-102, the sensor device or iohexol. Injection site reactions (bruising, erythema, extravasation) were also not considered related to MB-102.

A pivotal trial (protocol 100-003) enrolled 249 subjects. There were 31 adverse events reported in 26 subjects (10.4%). All reported events are mild or moderate in severity. Only 1 event (moderate nausea) was considered related to MB-102. No severe or serious events have been reported.

There may also be other risks that are unforeseen at this time. For additional information on the risk profile, please reference the current Investigator's Brochure.

# 8.2 MediBeacon® Transdermal GFR Measurement System

There are no direct risks associated with the MediBeacon<sup>®</sup> Transdermal GFR Measurement System (monitor portion) as it does not contact the study subject. Adverse events observed from the sensors are with regard to the methods used to affix it to the study subject. Risks may include a reaction to the sensor or adhesive material or the adhesive used on the skin clip.

## 8.2.1 Adhesive Clip

As with the adhesive used on the sensors, there is the chance of reaction to the adhesive used to attach the clip to the skin. Reactions could include redness, itchiness or other localized skin reactions. Clips will be provided, however other means (surgical tape, tegaderm, etc.) to secure the sensor cord may be used.

#### 8.3 Trial Procedures

Blood collection may lead to light-headedness and dizziness in some study subjects. It is recommended to ensure subjects continue to hydrate and eat during the dosing day to mitigate the effect of blood loss.

Bruising and pain at the site of the venous catheters may also be expected.

#### **8.3.1** Dose Extravasations

Should a dosing extravasation occur, a subject may report pain or burning during the injection. Subjects should be queried during the injection regarding any sensation. Subjects with MB-102 or saline extravasations will be discontinued from PK collection and fluorescent measurements but continued in the study for safety. All extravasations will be collected as adverse events and protocol deviations.

#### 9 Statistical Methods

#### 9.1 Overview

The transdermal-derived GFR data (tGFR) is obtained directly from the MediBeacon<sup>®</sup> Transdermal GFR Measurement System (TGFR) for each subject. This tGFR value is compared to the subject's nGFR<sub>BSA</sub> for the study endpoint determination.

## 9.2 Analysis Populations

The following analysis populations will be defined for the study:

➤ Intent-to-Measure (ITM) Population – The ITM population will consist of all subjects who are enrolled in the study in Stratum 1 & 2 and for whom an average session tGFR or

\_\_\_\_\_\_

- an average snapshot tGFR\* has been calculated, and who have not had any major protocol deviations that would impact TGFR system performance.
- ➤ Modified Intent-to-Measure (mITM) Population The mITM population will consist of all subjects in the ITM population with no outlier PK parameters.
- > Safety Population The safety population will consist of all subjects who are enrolled in the study and have been dosed with MB-102.
- ➤ **Pharmacokinetic (PK) Population** The pharmacokinetic population will consist of all subjects who are enrolled in the study and have any PK data.
- \* Note: this includes short gaps in data that are less than 30 minutes due to a resumption of the monitoring session where an "average snapshot GFR" is reported instead of a "average session GFR".

The mITM population will be the primary analysis set for all effectiveness analyses. The Safety Population will be used for the analysis of all safety variables and baseline characteristics. The PK Population will be used for the analyses of PK data.

Note: Data from the Run-in Cohort and Validation Cohort 1 will be considered Tuning Data and will not be used in the final analyses.

## 9.3 Subject Disposition

The number and percentage of subjects who complete the study or who terminate early from the study and the reasons for early termination will be collected and reported. Subjects will be considered to have completed the study if they complete the dosing day.

The number and percentage of subjects in each analysis population will be presented. Percentages will be based on the number of subjects enrolled.

#### 9.4 Plasma Pharmacokinetic Analyses

The pharmacokinetic objective is to characterize the single dose pharmacokinetics of MB-102 following IV bolus dosing, specifically, to obtain the clearance and total volume of distribution of MB-102 using compartmental methods in Phoenix WinNonlin (Certara, Version 8.1 or higher).

Based on prior data, it is expected that a two-compartment model will adequately describe the pharmacokinetic profiles of MB-102. The following two-compartmental pharmacokinetic parameters will be determined:

- C<sub>max</sub>: The maximum plasma concentration.
- > AUC: Area under the plasma concentration-time curve
- ightharpoonup  $t_{1/2\alpha}$ : Half-life associated with distribution phase
- $\succ$  t<sub>1/26</sub>: Half-life associated with elimination phase
- $\succ$   $t_{1/2}$ : elimination half-life from central compartment.

- > V: Total volume of distribution
- > CL: Systemic clearance
- ➤ V1: Volume of distribution for central compartment
- > V2: Volume of distribution for peripheral compartment

The two key PK parameters from compartmental analysis are CL and V. The clearance (CL) derived from the two-compartment model is the plasma-derived GFR used to calculate the BSA indexed nGFR that is the comparison to the tGFR for the P30 calculations. V is used in the calculation of GFR indexed to volume of distribution.

All PK concentrations and parameters will be listed. As each subject will have a unique GFR measurement, summary statistics are not applicable in this analysis.

Individual figures will be provided for plasma PK concentrations. All figures will be produced on both linear-linear and logarithmic-linear scales with data and the two-compartment fit.

# 9.5 Primary Endpoint Analysis

The primary endpoint is the performance measure of P30 for transdermal-derived GFR with respect to the plasma-derived indexed GFR, with a 95% confidence interval. The performance goal is 85%. Success for the study will be that the lower limit of the 95% CI is greater than 85%.

Prior data demonstrated for a P30 true value of 0.95, alpha of 0.025, performance goal of 85%, power of 90%, the one-sided exact binomial test yields a sample size of 102. As the reusable sensor is new, an adaptive trial design will be employed.

A Run-in Cohort of up to 30 evaluable subjects will be enrolled to test monitor algorithm settings with the TGFR reusable sensor with disposable adhesive ring. Additional run-in subjects may be enrolled at new clinical sites to ensure protocol compliance. Run-in subject data will be considered tuning data. The following will be enrolled into the run-in cohort:

- o At least 5 subjects will be enrolled in Stratum 2
- o At least 4 subjects in each of the FSS I-II; III-IV and V-VI
- Validation Cohort 1 (approximately 20 evaluable subjects) will be used to confirm final algorithm selection. Validation Cohort 1 subject data will be considered tuning data.
- Validation Cohort 2 (approximately 75 evaluable subjects) will be analysed in an interim analysis to compare results against the primary endpoint specification. At that time, the primary endpoint null hypothesis will be tested using an exact binomial test at a one-sided nominal alpha level of 0.0150 using the method of Pocock for a two-stage design with the interim analysis performed based on the first 53.57% of the planned number of subjects. At the final analysis, the primary endpoint null hypothesis will also be tested at a one-sided nominal alpha level of 0.0150. This will control the overall Type I error rate at the one-sided 0.025 level.

- If the primary endpoint has been achieved, the study will be terminated. If not, the trial will be continued.
- Validation Cohort 3 (approximately 65 evaluable subjects) will be enrolled in the event the interim analysis did not meet the primary outcome measure. Final analysis will be of the 140 evaluable subjects.

## 9.6 Safety Analyses

Safety of MB-102 will be evaluated through treatment emergent adverse events (TEAEs), where treatment emergence is defined with respect to the first dose of MB-102.

Safety of the MediBeacon® Transdermal GFR Measurement System will be evaluated through TEAEs, where treatment emergence is defined with respect to the start time of Transdermal GFR Measurement System use (placement of the sensor on the skin).

Additional safety variables include physical examinations, clinical laboratory assessments, ECGs, and concomitant medication use.

All safety analyses will be done for subjects receiving a single dose of MB-102.

# 9.6.1 Treatment-Emergent Adverse Events

AEs will be coded using the *Medical Dictionary for Regulatory Activities* (MedDRA). The system organ class and preferred term for each AE will be available, along with the verbatim reported term, event start and stop dates/times, seriousness, severity, relationship to treatment/device, action taken, and event outcome. SAEs will also be documented in a case narrative format.

The overall numbers and percentages of subjects who experienced any treatment-emergent AEs (TEAEs) will be presented. TEAEs will also be summarized at the subject level by system organ class and preferred term, and at the event level by system organ class/preferred term and severity and by system organ class/ preferred term and relationship to treatment.

# 9.6.2 Physical Examinations/Limited Physical Assessments

The results of physical examinations will be collected as adverse events if clinically significant or as medical history (if observations are noted prior to TGFR start). Physical exam data will not be listed.

# 9.6.3 Clinical Laboratory Assessments

Clinical laboratory tests include clinical chemistry, hematology, urinalysis and coagulation parameters. Each parameter will be summarized using the descriptive statistics. Details will be specified in the Statistical Analysis Plan (SAP). Also, individual subject results will be assessed against an appropriate reference range if available. The manifestation of any clinically significant abnormality that develops during the study will be reported as an AE.

#### 9.6.4 ECGs

ECG data will be listed. Clinically significant findings noted after dosing will be noted as adverse events.

# 9.6.5 Prior and Concomitant Therapies

Concomitant medications administered within 3 days prior to MB-102 dose administration and through the follow-up study visit will be listed. Medications will be coded using the World Health Organization (WHO) drug dictionary. Data will be provided in one or more subject data listings. Concomitant non-drug therapies will be listed.

# 9.7 Determination of Sample Size

For a P30 true value of 0.95, alpha of 0.025, performance goal of 85%, power of 90%, the one-sided exact binomial test yields a sample size of 102.

#### 9.8 Missing Data

Missing values will not be imputed.

### 10 Quality Assurance and Quality Control

## 10.1 Training

The clinical site will be trained on the protocol and study procedures. In addition, Sponsor representatives may be onsite during dosing procedures for the initial subjects at each site to assist sites with the operation of the MediBeacon® Transdermal GFR Measurement System.

#### 10.2 Audit and Inspection

The study site and study documentation may be subject to quality assurance audits during the course of the study by the sponsor, or its nominated representative. In addition, inspections may be conducted by regulatory authorities at their discretion.

## 10.3 Monitoring

Data for each subject will be recorded in an electronic data capture (EDC) system. Data collection must be completed for each subject enrolled in the study.

In accordance with GCP and International Council on Harmonization (ICH) guidelines, the study monitor will conduct monitoring visits at regular intervals. During the visits, the study monitor will perform the source document verification and verification that investigator's obligations and all applicable regulatory requirements are being fulfilled. The frequency of monitoring visits will be determined by the rate of subject recruitment.

The investigator must permit the monitor, the IEC, the sponsor's internal auditors and representatives from regulatory authorities direct access to all study-related documents and pertinent hospital or medical records, including direct access to electronic medical records for confirmation of data contained within the EDC system. Subject confidentiality will be protected at all times.

## 10.4 Data Management and Coding

MediBeacon or designee will be responsible for activities associated with the data management of this study. This will include setting up a relevant database and data transfer mechanisms, along with appropriate validation of data and resolution of queries. Data generated within this clinical study will be handled according to the relevant SOPs at MediBeacon or their designee.

Study sites will enter data into a 21 CFR Part 11 compliant electronic data capture (EDC) system via a secure internet connection. Data entered into the EDC system must be verifiable against source documents at the study site. Any changes to the data entered into EDC system will be recorded in the audit trail

Missing or inconsistent data will be queried via the EDC system to the investigator for clarification. Subsequent modifications to the database will be documented.

Fluorescent data from the TGFR System will be downloaded to hard media then transferred electronically to the Data Management designee via a secure data transfer process per the Study Procedure Manual.

All medical terms (medical history, concomitant medications and adverse events) will be coded.

#### 10.5 Protocol Deviations

The Investigator will not deviate from the clinical protocol without the prior written approval of MediBeacon except in medical emergencies or in unforeseen, isolated instances where minor changes are made that will not increase the subject's risk or affect the validity of the study. In medical emergencies, prior written approval for protocol deviations will not be required, but MediBeacon or their designee must be notified via telephone within 24 hours of occurrence. Prospective approval of protocol deviations to recruitment and enrolment criteria (also known as protocol waivers or exemptions) are not permitted.

Major Protocol Deviation is a significant deviation from the protocol that may impact subject safety and/or affect the integrity of clinical trial data. These may include, but are not limited to the following:

- Improper or inadequate informed consent procedures
- Subject did not meet eligibility criteria
- Subject received prohibited concomitant medication(s) at any time during the trial
- A significant protocol required assessment or procedure was not performed per protocol requirements

- Subject received incorrect study medications at any time during the trial
- Significant departure from protocol-required dosing (dosing extravasation)
- Subject developed criteria that required withdrawal from study protocol but was not withdrawn
- The sensor was removed prior to measurement of a tGFR
- An Average Session GFR or an Average Snapshot GFR was not obtained
- Sensors that are not cleaned and disinfected between study subjects

A Minor Protocol Deviation is a deviation that does not impact subject safety and/or compromise the integrity of the clinical trial data.

Subjects who experience a sensor dislodgement, a dosing or device issue or an extravasation (which would be considered a major deviation) will have PK sample collection discontinued and the sensor removed, but will be asked to remain in the study for safety follow-up (including dosing day safety assessments and the follow-up visit). The event that triggered the discontinuation of PK / fluorescent data collection will be considered the protocol deviation, however missing PK sample collections will not need to be documented as individual protocol deviations.

Deviations will be documented at the site and submitted to the IEC (as required) and the sponsor.

#### 10.6 Direct Data Collection

Fluorescent measurements will be collected directly by the MediBeacon<sup>®</sup> Transdermal GFR Measurement System and will not appear on any available source documentation with the exception of the tGFR which will be recorded onto the site source document and transcribed into the EDC. The MediBeacon<sup>®</sup> Transdermal GFR Measurement System will be a closed system.

#### 11 Records / Retention

Essential documents are those documents that individually and collectively permit evaluation of the study and quality of the data produced. After completion of the study, all documents and data relating to the study will be kept in an orderly manner by the investigator in a secure study file. All study records will be available for inspection by the sponsor or its representatives, or a regulatory agency.

Investigator files containing all records and reports of the investigation should be retained for a minimum of two (2) years (US) after the completion/ termination of the investigational study or the date that the records are no longer required for purposed of supporting a premarket approval application. The Sponsor will determine with the investigational site as to this exact date so that the minimum two-year record retention can be accomplished. Records may be discarded upon written notification by the Sponsor. To avoid error, the Principal Investigator should contact MediBeacon, before the destruction of any records and reports pertaining to the study to ensure they no longer need to be retained.

In addition, in accordance with the Clinical Trial Agreement, the Sponsor should be contacted if

the Principal Investigator plans to leave the investigational site so that appropriate arrangements for file custodianship can be made.

The following records must be maintained in designated study administrative files:

- Clinical protocol and all amendments
- Signed Investigator Agreement
- Independent Ethics Committee Approval Letter(s)documenting review and approval of all protocols, amendments, IBs, ICFs, subject materials, etc.
- IEC-approved informed consent(s) (including any revisions)
- Current CV for all Investigators and subinvestigators including evidence of current medical licensure
- Financial Disclosure Form for all Investigators
- Site Delegation of Authority Log
- Correspondence relating to this study
- Correspondence with the IEC
- IEC membership list and/or assurance
- Investigational site authorized study personnel signature list and delegation of authority
- Device Instructions for Use
- Lab certification, including a set of the lab's normal range for tests performed
- EDC Completion Guidelines
- Subject Screening & Enrolment Log
- Site Visit Log (e.g. for Monitor sign-in)
- Site Training records
- Investigational Device and Drug Accountability Logs
- Reports (includes Adverse Event reports and final reports from Investigator and Sponsor)
- Copy of all EC approved subject-related materials and/or study advertising materials

The following records must be maintained for each subject enrolled in the study:

- Signed subject consent forms
- Electronic copy of final completed case reports (to be provided by the sponsor at the end of the study)
- Jump drive with subject's fluorescent data from the TGFR system
- All lab work and testing results
- Record of any complications, adverse events, device problems and/or malfunctions, with supporting documentation
- Procedure reports, progress notes, physician and/or nursing notes, and subject office files
- Records pertaining to subject deaths

#### 12 Ethics

## 12.1 Independent Ethics Committee (IEC)

Before initiation of the study at each study site, the protocol, all protocol amendments, Investigator's Brochure, the ICF, the subject information sheet and any other relevant study documentation will be submitted to the appropriate IEC. Written approval of the study and all relevant study information must be obtained before the study site can be initiated or the study device is released to the investigator. Any necessary extensions or renewals of IEC approval must be obtained, in particular, for changes to the study such as modification of the protocol, the ICF, the written information provided to subjects, and/or other procedures.

The investigator will report promptly to the IEC any new information that may adversely affect the safety of the subjects or the conduct of the study. The investigator will submit written summaries of the study status to the IEC annually, or more frequently if requested by the IEC. On completion of the study, the site will notify the IEC that the study has ended.

## 12.2 Ethical Conduct of the Study

The ICH guidelines for current GCP (ICH R2, 2016), the Code of Federal Regulations Title 21 CFR Parts 812, 11, 50, 54 and 56 and ISO 14155: 2020(E) Clinical Investigation of Medical Devices for Human Subjects – Good Clinical Practice, as well as the ethical principles defined by the World Medical Association Declaration of Helsinki, and the requirements of national device and data protection laws and other applicable regulatory requirements will be followed.

## 12.3 Subject Information and Consent

The investigator is responsible for ensuring that no subject undergoes any study related examination or activity before that subject has given written informed consent to participate in the study. The written consent must be given by the subject, after detailed information about the study has been given and in accordance with any national provisions on the protection of clinical study subjects. The verbal explanation will cover all the elements specified in the written information provided for the subject.

The investigator or designated personnel will inform the subject of the objectives, methods, anticipated benefits, and potential risks and inconveniences of the study. The subject should be given every opportunity to ask for clarification of any points he/she does not understand and, if necessary, ask for more information. At the end of the interview, the subject will be given time to consider the study, if this is required, or if the subject requests more time. Subjects and/or legally authorized representatives will be required to sign and date the ICF. After signatures are obtained, a copy will be provided to the subject, and a signed ICF will be kept and archived by the investigator in the investigator's study file for possible inspection by regulatory authorities, the IEC, or sponsor.

It should be emphasized to the subject that he/she is at liberty to withdraw from the study at any time, without penalty or loss of benefits to which the subject is otherwise entitled. Subjects who

refuse to give or who withdraw written informed consent should not be included or continue in the study.

## 12.4 Financing and Insurance

This clinical trial will be sponsored by MediBeacon and its conduct will be governed under an executed Clinical Trial Agreement that will define the coverage of costs associated with study implementation by the trial site. MediBeacon will maintain appropriate clinical trial insurance at limits agreed upon in the agreement.

## 12.5 Subject Confidentiality

All personal data collected and processed for the purposes of this study should be managed by the investigator and his/her staff with adequate precautions to ensure confidentiality of those data, in accordance with applicable national and/or local laws and regulations on personal data protection.

Monitors, auditors, and other authorized agents of the sponsor and/or its designee, the ethics committees approving this research, and any other applicable regulatory agency(ies), will be granted direct access to the study subjects' original medical records (including electronic medical records) for verification of clinical study procedures and/or data, without violating the confidentiality of the subjects to the extent permitted by the law and regulations. In any presentations of the results of this study or in publications, the subjects' identity will remain confidential.

#### 12.6 Reporting and Publication, Including Archiving

Publication of all study results in the form of abstracts, manuscripts, presentations, posters, etc. will be developed in accordance with the Clinical Trial Agreement.

#### 13 References

Agarwal R. Ambulatory GFR measurement with cold iothalamate in adults with chronic kidney disease. Am J Kidney Dis. 2003 Apr; 41(4): 752-9.

Endre ZH, Pickering JW, Walker RJ. Clearance and beyond: the complementary roles of GFR measurement and injury biomarkers in acute kidney injury (AKI). Am J Physiol Renal Physiol 2011 301: F697-F707.

Erley CM, Bader BD, Berger ED, et al. Plasma clearance of iodine contrast media as a measure of glomerular filtration rate in critically ill patients. Crit Care Med. 2001 Aug; 29(8):1544-50.

Fitzpatrick TB. Soleil et peau [Sun and skin]. Journal de Médecine Esthétique. 1975; 2:33-34

Kidney Disease Statistics for the United States. http://kidney.niddk.nih.gov/kudiseases/pubs/kustats/index.aspx#13

Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A New Equation to Estimate Glomerular Filtration Rate. Ann Intern Med. 2009 May 5;150(9):604-12.

National Institutes of Health Web Site (Bethesda MD, 08 October 2008), "Annual report targets chronic kidney disease in the United States," http://www.nih.gov/news/health/oct2008/niddk-08.htm

Stevens, LA and Levey, AS. Measured GFR as a Confirmatory Test for Estimated GFR. 2009. J. Am Soc Nephrol 20: 2305-2313.

Stevens LA, Coresh J, Greene T, Levey AS. Assessing kidney function--measured and estimated glomerular filtration rate. N Engl J Med. 2006 Jun 8;354 (23):2473-83.

Verhave JC, Fesler P, Ribstein J, du Cailar G, Mimran A. Estimation of renal function in subjects with normal serum creatinine levels: influence of age and body mass index. Am J Kidney Dis. 2005 Aug; 46(2): 233-41.

# 14 Appendix A Fitzpatrick Scale

The Fitzpatrick Scale (shown below) will be determined via measurements of melanin using the Mexameter on the upper chest area where the sensor is anticipated to be placed. As a general reference, the subjective skin color scale is show below.

# The Fitzpatrick Scale



Source: Fitzpatrick, 1975

Mexameter melanin measurements correspond to FSS scores as noted below:

| 0 | FSS type I: | Mexameter melanin range: | 0 - 100 |
|---|---------------|--------------------------|-----------|
| 0 | FSS type II: | Mexameter melanin range: | 100 - 150 |
| 0 | FSS type III: | Mexameter melanin range: | 150 - 250 |
| 0 | FSS type IV: | Mexameter melanin range: | 250 - 350 |
| 0 | FSS type V: | Mexameter melanin range: | 350-450 |
| 0 | FSS type VI: | Mexameter melanin range: | 450 - 999 |

## **Investigator Signature Page**

**Protocol Title:** An Open Label, Multi-Center, Safety and Pharmacokinetic

Bridging Study of MB-102 (Relmapirazin) and the Use of the MediBeacon<sup>®</sup> Transdermal GFR Measurement System using the TGFR Reusable Sensor with Disposable Adhesive Ring in Normal and Renal Compromised Subjects for the Evaluation of Kidney

**Function** 

**Protocol Number:** 100-201

## Confidentiality and cGCP Compliance Statement

I, the undersigned, have reviewed this protocol, including appendices and other documents that may be considered part of the investigational plan, and I will conduct the study as described in compliance with this protocol, GCP, the ethical principles defined by the World Medical Association Declaration of Helsinki (2013), applicable regional regulations and relevant ICH guidelines.

Once the protocol has been approved by the IEC, I will not modify this protocol without obtaining prior approval of the MediBeacon Inc. and of the IEC. I will submit the protocol modifications and/or any ICF modifications to MediBeacon Inc. and IEC, and approval will be obtained before any modifications are implemented.

I understand that all information obtained during the conduct of the study with regard to the subjects' state of health will be regarded as confidential. No subjects' names will be disclosed. All subjects will be identified by assigned numbers on all eCRFs, laboratory samples or source documents forwarded to the sponsor. Clinical information may be reviewed by the sponsor or its agents or regulatory agencies. Agreement must be obtained from the subject before disclosure of subject information to a third party.

I will oversee all aspects of study conduct and will only appropriately delegate responsibilities to adequately qualified and trained staff. I will oversee the completion of source data collection such that all data collected for the study may be substantiated against accurate source medical records.

| Information developed in this clinical study may clinical investigators, regulatory agencies, or othe required. | |
|---|---|
| Investigator Signature | Date |

# 15 Signature of the Sponsor's Responsible Officers

#### 15.1 Chief Scientific Officer

Richard Dorshow, PhD

MediBeacon Inc. 425 N. New Ballas Road St. Louis, MO 63141 USA

#### 15.2 Medical Officer

Dr. Joseph Pierro

MediBeacon Inc. 425 N. New Ballas Road St. Louis, MO 63141 USA

Phone: (Central Time; United States)